CLINICAL TRIAL: NCT04338321
Title: A Randomized, Open-label, Rater-Blinded, Active-Controlled, International, Multicenter Study to Evaluate the Efficacy, Safety, and Tolerability of Flexibly Dosed Esketamine Nasal Spray Compared With Quetiapine Extended-Release in Adult and Elderly Participants With Treatment-Resistant Major Depressive Disorder Who Are Continuing a Selective Serotonin Reuptake Inhibitor/Serotonin-Norepinephrine Reuptake Inhibitor
Brief Title: A Long-term Comparison of Esketamine Nasal Spray Versus Quetiapine Extended Release, Both in Combination With a Selective Serotonin Reuptake Inhibitor/Serotonin-Norepinephrine Reuptake Inhibitor, in Participants With Treatment Resistant Major Depressive Disorder
Acronym: ESCAPE-TRD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen-Cilag International NV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR108787; 2019-002992-33 (EudraCT Number); 54135419TRD3013 (Other: Janssen-Cilag International NV)
Record Dates: First submitted 2020-04-06; First posted 2020-04-08 (Actual); Results first posted 2023-02-15 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Esketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Esketamine Arm (Experimental): Participants will receive treatment with esketamine nasal spray (28 milligram [mg] [initial dose for elderly participants 65 to 74 years of age and adults of Japanese ancestry; may be used throughout the study in these populations; may be uptitrated in 28 mg increments], 56 mg [initial dose for adult participants aged 18 to 64 years and may be used for all age groups throughout the study], or 84 mg [maximum dose esketamine nasal spray may be uptitrated to]) twice-weekly with a flexible dose regimen from Day 1 until Week 4, once weekly from Week 5 to Week 8 and once-weekly or once every 2 weeks from Week 9 to Week 32 in combination with continuing serotonin-norepinephrine reuptake inhibitor/selective serotonin reuptake inhibitor (SSRI/SNRI).
  Interventions: Drug: Esketamine 28 mg; Drug: Esketamine 56 mg; Drug: Esketamine 84 mg; Drug: SSRI/SNRI
- Comparator Arm (Active Comparator): Participants will continue to take their current SSRI/SNRI augmented with quetiapine extended release (XR) as per the Summary of Product Characteristics (SmPC) (or local equivalent, if applicable). In adult participants aged 18 to 64 years, the initial dose is 50 mg/day on Days 1-2, 150 mg/day on Days 3-4 [lowest effective dose]; a further dose increase to 300 mg/day on Day 5 and onward will be based on individual participant evaluation. In elderly participants aged 65 to 74 years, the initial dose is 50 mg/day on Days 1-3, 100 mg/day on Days 4-7, and 150 mg/day on Day 8; a further dose increase to 300 mg/day will be based on individual participant evaluation no earlier than Day 22.
  Interventions: Drug: Quetiapine XR 50 mg; Drug: Quetiapine XR 100 mg; Drug: Quetiapine XR 150 mg; Drug: SSRI/SNRI

INTERVENTIONS:
Drug: Esketamine 28 mg — Esketamine will be self-administered at a dose of 28 mg as nasal spray.
  Arms: Esketamine Arm
Drug: Esketamine 56 mg — Esketamine will be self-administered at a dose of 56 mg as nasal spray.
  Arms: Esketamine Arm
Drug: Esketamine 84 mg — Esketamine will be self-administered at a dose of 84 mg (maximum uptitrated dose) as nasal spray.
  Arms: Esketamine Arm
Drug: Quetiapine XR 50 mg — Quetiapine XR will be administered at an initial dose of 50 mg/day and may be further increased to 300 mg/day based on individual participant evaluation.
  Arms: Comparator Arm
Drug: Quetiapine XR 100 mg — Quetiapine XR will be administered at a dose of 100 mg/day and may be further increased to 300 mg/day based on individual participant evaluation.
  Arms: Comparator Arm
Drug: Quetiapine XR 150 mg — Quetiapine XR will be administered at a dose of 150 mg/day and may be further increased to 300 mg/day based on individual participant evaluation.
  Arms: Comparator Arm
Drug: SSRI/SNRI — Participants will continue to take SSRI/SNRI that is approved for use in depression in their country of participation; off-label use of any SSRI/SNRI is not permitted. The continuing SSRI/SNRI dosage may be optimized throughout the study, at the investigator's discretion and based on the SmPC (or local equivalent, if applicable).

SUMMARY:
The primary purpose of this study is to evaluate the efficacy of flexibly dosed esketamine nasal spray compared with quetiapine extended-release (XR), both in combination with a continuing selective serotonin reuptake inhibitor/serotonin-norepinephrine reuptake inhibitor (SSRI/SNRI), in achieving remission in participants who have treatment-resistant major depressive disorder (MDD) with a current moderate to severe depressive episode.

DETAILED DESCRIPTION:
A depressive state with classical symptoms such as low (depressive/sad) mood, markedly diminished interest in activities, significant weight loss/gain, insomnia or hypersomnia, psychomotor agitation/retardation, excessive fatigue, inappropriate guilt, diminished concentration, and recurrent thoughts of death, persisting for more than 2 weeks is classified as major depressive disorder (MDD). The mechanism of action of ketamine is distinct from conventional antidepressants (ADs), which target the monoamines (serotonin, norepinephrine, and/or dopamine). Esketamine, the S-enantiomer of ketamine, is approved and widely used for the induction and maintenance of anesthesia via intramuscular or intravenous (IV) administration. There is a significant unmet need to develop novel AD treatments based on the relevant psychophysiological pathways underlying MDD. The goal of any novel treatment would be the rapid and long-lasting relief of depressive symptoms, especially in participants with treatment-resistant depression (TRD), who lack a sufficient response to the currently available treatment strategies. The study consists of a Screening Phase (up to 14 days), an Acute Phase (8 Weeks), a Maintenance Phase (24 Weeks) and a Safety Follow-up Phase (2 Weeks). Safety assessment includes adverse event, serious adverse events, physical examination, vital signs, electrocardiogram, clinical safety laboratory assessments, suicidal risk monitoring. The total duration of the study is approximately 36 Weeks for all participants.

ELIGIBILITY:
Inclusion Criteria:

* At screening, each participant must meet Diagnostic and Statistical Manual of Mental Disorders, fifth edition (DSM-5) diagnostic criteria for single-episode major depressive disorder (MDD) or recurrent MDD, without psychotic features, based on clinical assessment and confirmed by the Mini International Neuropsychiatric Interview (MINI)
* At screening and baseline, each participant must have an Inventory of Depressive Symptomatology - Clinician-rated, 30 item (IDS-C30) total score of greater than or equal to (>=) 34
* Must be on a current antidepressive treatment that includes an selective serotonin reuptake inhibitor (SSRI)/ serotonin-norepinephrine reuptake inhibitor (SNRI) at screening that resulted in nonresponse (less than 25% improvement of symptoms) after having been given at an adequate dosage (based on antidepressive dosages from SmPC [or local equivalent, if applicable]) for an adequate duration of at least 6 weeks and having been uptitrated to the maximum tolerated dose; however, at screening the participant must show signs of minimal clinical improvement to be eligible for the study. Clinical improvement of a participant on their current AD treatment will be retrospectively evaluated in a qualified psychiatric interview performed by an experienced clinician. At baseline (Day 1) prior to randomization, the investigator will evaluate any changes in the participant's signs/symptoms of depression since the screening assessment and confirm that the inclusion criteria for the current AD treatment are still met (that is nonresponse and minimal clinical improvement)
* The current antidepressive treatment, was immediately preceded by nonresponse to at least 1 but not more than 5 different, consecutive treatments (all within the current moderate to severe antidepressive episode) with anti-depressants (ADs) taken at an adequate dosage for an adequate duration of at least 6 weeks and must be documented
* Must have been treated with at least 2 different antidepressive substance classes among the treatments taken at an adequate dosage for an adequate duration of at least 6 weeks resulting in nonresponse in the current moderate to severe depressive episode (including the current treatment with an selective serotonin reuptake inhibitor/serotonin-norepinephrine reuptake inhibitor [SSRI/SNRI])
* Must be on a single oral SSRI/SNRI on Day 1 prior to randomization

Exclusion Criteria:

* Received treatment with esketamine or ketamine in the current moderate to severe depressive episode
* Received treatment with quetiapine extended- or immediate-release in the current moderate to severe depressive episode of a dose higher than 50 milligram per day (mg/day)
* Had depressive symptoms in the current moderate to severe depressive episode that previously did not respond to an adequate course of treatment with electroconvulsive therapy (ECT), defined as at least 7 treatments with unilateral/bilateral ECT
* Has no signs of clinical improvement at all or with a significant improvement on their current AD treatment that includes an SSRI/SNRI as determined at screening by an experienced clinician during the qualified psychiatric interview
* Received vagal nerve stimulation or has received deep brain stimulation in the current episode of depression
* has a current or prior DSM-5 diagnosis of a psychotic disorder or MDD with psychotic features, bipolar or related disorders (confirmed by the Mini International Neuropsychiatric Interview [MINI]), obsessive compulsive disorder (current only), intellectual disability (DSM-5 diagnostic codes 317, 318.0, 318.1, 318.2, 315.8, and 319), autism spectrum disorder, borderline personality disorder, or antisocial personality disorder, histrionic personality disorder, or narcissistic personality disorder
* age at onset of first episode of MDD was more than or equal to (>=) 55 years
* has homicidal ideation or intent, per the investigator's clinical judgment; or has suicidal ideation with some intent to act within 1 month prior to screening, per the investigator's clinical judgment; or based on the Columbia-Suicide Severity Rating Scale (C-SSRS), corresponding to a response of "Yes" on Item 4 (active suicidal ideation with some intent to act, without specific plan) or Item 5 (active suicidal ideation with specific plan and intent) for suicidal ideation, or a history of suicidal behavior within the past year prior to screening. Participants reporting suicidal ideation with intent to act or suicidal behavior prior to the start of the acute phase should also be excluded

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 676 (Actual)
Dates: Start 2020-08-21 (Actual); Primary Completion 2022-01-20 (Actual); Study Completion 2022-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen-Cilag International NV Clinical Trials, Study Director — Janssen-Cilag International NV
Locations (171):
- Argentina (8):
  - Fundacion para el Estudio y Tratamiento de las Enfermedades Mentales, Buenos Aires
  - FunDaMos, Buenos Aires
  - CEN Consultorios Especializados en Neurociencias, Córdoba
  - Fundacion Lennox, Córdoba
  - Instituto Medico DAMIC, Córdoba
  - Sanatorio Prof Leon S Morra S A, Córdoba
  - Instituto de Neurociencias San Agustin, La Plata
  - C I A P Centro de investigacion y Asistencia en Psiquiatria, Rosario
- Austria (3):
  - Medical University Graz, Graz
  - Schmitz and Schmitz, Vienna
  - Medical University Vienna MUV, Vienna
- Belgium (6):
  - Anima, Alken
  - Pz Duffel, Duffel
  - Clinique Psychiatrique des Frères Alexiens, Henri-Chapelle
  - Sint-Franciskusziekenhuis, Heusden-Zolder
  - ARIADNE, Lede
  - CHU de Liege, Liège
- Brazil (5):
  - CPN - Centro de Pesquisa em Neurociências Ltda, Belo Horizonte
  - Trial Tech Tecnologia em Pesquisas com Medicamentos, Curitiba
  - Ruschel Medicina e Pesquisa Clínica Ltda, Rio de Janeiro
  - C J S Carvalho & Carvalho LTDA (Viver - Centro De Desospitalizacao Humana), São Paulo
  - BR Trials, São Paulo
- Bulgaria (8):
  - State Psychiatric Hospital Kardzhali, Kardzhali
  - UMHAT 'Dr. Georgi Stranski', EAD, Pleven
  - Mental Health Center - Plovdiv, Plovdiv
  - Mental Health Center - Rousse, Rousse
  - Multiprofile Hospital for Active Treatment in Neurology and Psychiatry Sveti Naum, Sofia
  - MHC - Sofia, EOOD, Sofia
  - Centre for Mental Health Prof.N.Shipkovenski EOOD, Sofia
  - University Multiprofile Hospital for Active Treatment - UMHAT Alexandrovska EAD, Sofia
- Czechia (8):
  - Psychiatricka ambulance Saint Anne s.r.o., Brno
  - Psychiatricka ambulance, MUDr. Marta Holanova, Brno
  - NeuropsychiatrieHK, s.r.o., Hradec Kralove-Vekose
  - A Shine S R O, Pilsen
  - Clintrial s r o, Prague
  - AD71 s.r.o., Prague
  - Medical Services Prague S R O, Prague
  - Institut Neuropsychiatricke pece, Prague
- Denmark (2):
  - Aalborg University Hospital, Aalborg
  - Psykiatrien i Region Syddanmark, Esbjerg N
- Finland (3):
  - Mederon LTD at ARTES, Helsinki
  - Psykiatrinen Palvelukeskus Solvum Oy, Helsinki
  - Savon Psykiatripalvelu, Kuopio
- Germany (38):
  - Universitaetsklinikum der RWTH Aachen, Aachen
  - Rheinhessen Fachklinik Alzey, Alzey
  - Emovis GmbH, Berlin
  - Charite Campus Benjamin Franklin, Berlin
  - Medizinisches Versorgungszentrum LiO GmbH, Berlin
  - Alexander Schulze - Germany, Berlin
  - Praxis Dr. med. Kirsten Hahn, Berlin
  - Vivantes Klinikum Spandau, Berlin
  - Universitatsklinikum Bonn, Bonn
  - Klinikum Chemnitz gGmbH, Chemnitz
  - Carl-Thiem-Klinikum Cottbus gGmbH, Cottbus
  - Klinikum Dortmund gGmbH, Dortmund
  - Universitatsklinikum Carl Gustav Carcus Dresden, Dresden
  - Universitatsklinikum Frankfurt, Frankfurt am Main
  - Universitätsklinikum Freiburg - Abteilung für Psychiatrie u. Psychotherapie mit Poliklinik, Freiburg im Breisgau
  - SRH Waldklinikum Gera GmbH, Gera
  - Georg August Universitat Universitatsmedizin Gottingen, Göttingen
  - Evangelisches Krankenhaus Bethanien gGmbH, Greifswald
  - Universitaetsklinik Hamburg-Eppendorf, Hamburg
  - Klinische Forschung Hamburg, Hamburg
  - Klinische Forschung Hannover-Mitte GmbH, Hanover
  - Medizinische Hochschule Hannover, Hanover
  - Universität Heidelberg, Heidelberg
  - Oberhavel Kliniken GmbH, Hennigsdorf
  - Universitätsklinikum des Saarlandes, Homburg
  - Universitatsklinikum Jena, Jena
  - Panakeia - Arzneimittelforschung GmbH, Leipzig
  - Universitaetsklinikum Magdeburg A.oe.R, Magdeburg
  - Universitatsmedizin der Johannes Gutenberg Universitat Mainz, Mainz
  - Pharmakologisches Studienzentrum Chemnitz GmbH, Mittweida
  - Universitatsklinikum Munster, Münster
  - Ruppiner Kliniken, Neuruppin
  - Praxis Prof. Steinwachs, Nuremberg
  - Johanniter Krankenhaus Oberhausen, Oberhausen
  - Danuvius Klinik Pfaffenhofen Fachklinik für Psychiatrie, Psychotherapie und Psychosomatik, Pfaffenhofen
  - Somni Bene GmbH, Schwerin
  - Klinische Forschung Schwerin GmbH, Schwerin
  - Klinikum der Hansestadt Stralsund GmbH-Ambulanz-Klinik für Psychiatrie und Psychotherapie - Germany, Stralsund
- Greece (9):
  - Aiginition Hospital of Athens, Athens
  - 'Dafni' Psychiatric Hospital of Attica, Athens
  - Venizeleio General Hospital, Crete
  - Psychiatric Clinic 'Agios Charalampos', Heraklion
  - University General Hospital of Ioannina, Ioannina
  - University General Hospital of Rio Patras, Pátrai
  - 424 Military Hospital of Thessaloniki, Thessaloniki
  - Psychiatric Hospital of Thessaloniki, Thessaloniki
  - G Papanikolaou Hospital of Thessaloniki, Thessaloniki
- Hungary (9):
  - Semmelweis Egyetem, Budapest
  - Eszak Kozep budai Centrum Uj Szent Janos Korhaz es Szakrendelo Budai Csaladkozpontu, Budapest
  - Processus Kft, Budapest
  - Debreceni Egyetem, Kenézy Gyula Egyetemi Oktatókórház, Debrecen
  - Bugat Pal Korhaz, Gyöngyös
  - Petz Aladar Megyei Oktato Korhaz, Győr
  - Bács-Kiskun Megyei Kórház a Szegedi Tudományegyetem Általános Orvostudományi Kar Oktató Kórháza, Kalocsa
  - Szabolcs-Szatmar-Bereg Megyei Korhazak es Egyetemi Oktatokorhaz, Nyíregyháza
  - Pecsi Tudomanyegyetem Klinikai Kozpont, Pécs
- Israel (6):
  - Rambam Medical Center, Haifa
  - Shalvata Mental Health Center, Hod HaSharon
  - Beer Yaakov Mental Health Center, Lod
  - Geha Mental Health Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - Tel Aviv Sourasky Medical Center, Telaviv
- Kazakhstan (3):
  - Republican Scientific and Practical Center of Mental Health, Almaty
  - Medical Center for Psychological Healt SME, Nur-Sultan
  - East-Kazakhstan Regional Centre of Mental Health, Ust-Kamenogorsk
- Malaysia (5):
  - Hospital Raja Permaisuri Bainun, Ipoh
  - Hospital Kuala Lumpur, Kuala Lumpur
  - University Malaya Medical Centre, Kuala Lumpur
  - Hospital Pengajar Universiti Putra Malaysia, Serdang
  - Hospital Tuanku Jaafar, Seremban
- Netherlands (3):
  - Brain Research Center, Amsterdam
  - AMC, Amsterdam
  - LUMC, Leiden
- Norway (3):
  - Haukeland University Hospital, Hordaland
  - Sykehuset Ostfold, Moss
  - St Olav University Hospital, Trondheim
- Poland (10):
  - Mlynowamed Specjalistyczny Psychiatryczny Gabinet Lekarski Joanna Lazarczyk, Bialystok
  - Osrodek Badan Klinicznych CLINSANTE S C, Bydgoszcz
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - Centrum Badan Klinicznych PI House sp z o o, Gdansk
  - Centrum Medyczne Care Clinic Katowice, Katowice
  - Niepubliczny Zaklad Opieki Psychiatrycznej MENTIS, Leszno
  - Specjalistyczny Psychiatryczny Zespol Opieki Zdrowotnej w Lodzi Szpital im. J. Babinskiego, Lodz
  - SPZOZ CSK UM w Lodzi Klinika Zaburzen Afektywnych i Psychotycznych, Lodz
  - Centrum Medyczne Luxmed Sp z o o, Lublin
  - Osrodek Badan Klinicznych CLINSANTE S C, Torun
- Portugal (6):
  - Hospital de Braga, Braga
  - Centro Hospitalar do Tâmega e Sousa, EPE - Hospital Padre Americo, Vale do Sousa, Guilhufe - Penafiel
  - Hosp. Cuf Tejo, Lisbon
  - Fund. Champalimaud, Lisbon
  - Centro Hospitalar de Lisboa Norte Hospital Santa Maria, Lisbon
  - Uls Loures Odivelas - Hosp. Loures, Loures
- South Africa (3):
  - Cape Town Clinical Research Centre, Cape Town
  - Flexivest 14 Research, Cape Town
  - Gert Bosch Pretoria South Africa, Garsfontein
- South Korea (6):
  - Chonnam National University Hospital, Gwangju
  - Wonkwang University Hospital, Iksan
  - KyungHee University Hospital, Seoul
  - Korea University Anam Hospital, Seoul
  - Severance Hospital Yonsei University Health System, Seoul
  - Samsung Medical Center, Seoul
- Sweden (6):
  - Psykiatriska kliniken, Gothenburg
  - Affecta Pskyiatrimottagning, Halmstad
  - Psykiatriska kliniken, Luleå
  - ProbarE i Lund AB, Lund
  - ONE LIFETIME Lakarmottagning, Skövde
  - ProbarE i Stockholm AB, Stockholm
- Taiwan (10):
  - Changhua Christian Hospital, Changhua
  - Hualien Tzu Chi Hospital, Hualien City
  - Kai-Syuan Psychiatric Hospital, Kaohsiung City
  - Chang Gung Memorial Hospital, Kaohsiung City
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Mackay Memorial Hospital, Taipei
  - Taipei Medical University, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Chang Gung Memorial Hospital, Taoyuan District
- Turkey (Türkiye) (10):
  - Hacettepe University Medical Faculty, Ankara
  - Bursa Yuksek Ihtisas Training and Research Hospital, Bursa
  - Uludag University Medical Faculty, Bursa
  - Bakirkoy Mental Health Training and Research Hospital, Istanbul
  - Erenkoy Mental Health Hospital, Istanbul
  - Uskudar University Neuropsychiatry Hospital, Istanbul
  - Ege Universitesi Tip Fakultesi, Izmir
  - Selcuk University Medical Faculty, Konya
  - Liv Hospital, Samsun
  - Namik Kemal University, Tekirdağ
- American Center for Psychiatry and Neurology, Abu Dhabi, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale open Data Access (YODA) Project site at yoda.yale.edu
URL: https://www.janssen.com/clinical-trials/transparency

REFERENCES:
- [Derived] Lan CH, Wei JC. Esketamine Nasal Spray versus Quetiapine for Resistant Depression. N Engl J Med. 2024 Jan 4;390(1):93-94. doi: 10.1056/NEJMc2313230. No abstract available. PMID 38169503
- [Derived] Horowitz MA, Ploderl M, Naudet F. Esketamine Nasal Spray versus Quetiapine for Resistant Depression. N Engl J Med. 2024 Jan 4;390(1):93. doi: 10.1056/NEJMc2313230. No abstract available. PMID 38169502
- [Derived] Reif A, Bitter I, Buyze J, Cebulla K, Frey R, Fu DJ, Ito T, Kambarov Y, Llorca PM, Oliveira-Maia AJ, Messer T, Mulhern-Haughey S, Rive B, von Holt C, Young AH, Godinov Y; ESCAPE-TRD Investigators. Esketamine Nasal Spray versus Quetiapine for Treatment-Resistant Depression. N Engl J Med. 2023 Oct 5;389(14):1298-1309. doi: 10.1056/NEJMoa2304145. PMID 37792613

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who discontinued the treatment early still remained in the study and were followed up until the end of study.
Groups:
- Esketamine Nasal Spray + Oral Antidepressant (AD): Participants received treatment with esketamine nasal spray (28 milligrams [mg] [initial dose for elderly participants aged 65 to 74 years and adults of Japanese ancestry], 56 mg [initial dose for adult participants aged 18 to 64 years], or 84 mg [maximum dose esketamine nasal spray]) twice-weekly with a flexible dose regimen from Day 1 until Week 4, once weekly from Week 5 to Week 8 and once-weekly or once every 2 weeks from Week 9 to Week 32 in combination with continuing serotonin-norepinephrine reuptake inhibitor/selective serotonin reuptake inhibitor (SSRI/SNRI).
- Quetiapine Extended Release (XR) + Oral AD: Participants continued to take their current SSRI/SNRI augmented with quetiapine XR as per the Summary of Product Characteristics (SmPC) (or local equivalent, if applicable) at an initial dose of 50 mg/day on Days 1-2, 150 mg/day on Days 3-4 (lowest effective dose) in adult participants aged 18 to 64 years; a further dose increase to 300 mg/day on Day 5 and onward were based on individual participant evaluation. In elderly participants aged 65 to 74 years, the initial dose was 50 mg/day on Days 1-3, 100 mg/day on Days 4-7, and 150 mg/day on Day 8; a further dose increase to 300 mg/day were based on individual participant evaluation no earlier than Day 22.
Period: Overall Study
Arm/Group | Esketamine Nasal Spray + Oral Antidepressant (AD) | Quetiapine Extended Release (XR) + Oral AD
Started | 336 | 340
Treated (Safety Analysis Set) | 334 | 336
Completed Treatment | 258 | 203
Completed | 274 | 232
Not Completed | 62 | 108
Not completed — Adverse Event | 4 | 10
Not completed — Death | 1 | 1
Not completed — Lost to Follow-up | 4 | 9
Not completed — Withdrawal by Subject | 45 | 69
Not completed — Physician Decision | 5 | 9
Not completed — Other | 3 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Esketamine Nasal Spray + Oral Antidepressant (AD) | Quetiapine Extended Release (XR) + Oral AD | Total
Number analyzed (Participants) | 336 | 340 | 676
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.3 (13.6) | 45.7 (13.38) | 45 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 225 | 222 | 447
  Male | 111 | 118 | 229
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 9 | 10 | 19
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 7 | 12
  White | 137 | 152 | 289
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 185 | 171 | 356

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Remission as Assessed by the Montgomery-Asberg Depression Rating Scale (MADRS) Score at Week 8
Description: Percentage of participants with remission as assessed by the MADRS at Week 8 was reported. The MADRS is a clinician-rated scale designed to measure depression severity and to detect changes due to antidepressant treatment. The scale consists of 10 items, each of which is scored from 0 (item is not present or is normal) to 6 (severe or continuous presence of the symptoms), for a total possible score of 60. Higher scores represent a more severe condition. The MADRS evaluates apparent sadness, reported sadness, inner tension, sleep, appetite, concentration, lassitude, interest level, pessimistic thoughts, and suicidal thoughts. A participant was defined as being in remission if the MADRS total score was less than or equal to (<=)10 and no treatment or study discontinuation before Week 8.
Time Frame: Week 8
Population: The full analysis set (FAS) included all randomized participants.
Measure: Number; unit: Percentage of participants
Arm/Group | Esketamine Nasal Spray + Oral Antidepressant (AD) | Quetiapine Extended Release (XR) + Oral AD
Number analyzed (Participants) | 336 | 340
Percentage of participants | 27.1 | 17.6
Statistical Analysis 1: Comparison: Esketamine Nasal Spray + Oral Antidepressant (AD) vs Quetiapine Extended Release (XR) + Oral AD; Test type: Superiority; p = 0.003, Cochran-Mantel-Haenszel; Mean Difference (Final Values) = 9.44, 95% CI 2-sided [3.19 to 15.68]

2. Secondary Outcome: Percentage of Participants With Both Remission at Week 8 and Relapse-free Until Week 32
Description: Percentage of participants with both remission at Week 8 and relapse-free until Week 32 were reported. A participant was defined as being in remission if the MADRS total score was <= 10 and no treatment or study discontinuation before Week 8. A relapse was defined by any of following: a) Worsening of depressive symptoms as indicated by MADRS total score greater than or equal to (>=) 22 confirmed by 1 additional assessment of MADRS total score >= 22 within the next 5 to 15 days. The date of the second MADRS assessment was used for the date of relapse; b) Any psychiatric hospitalization for: worsening of depression, suicide prevention or suicide attempt, the start date of hospitalization was the date of relapse; c) Suicide attempt, completed suicide, or any other clinically relevant event determined by investigator's judgment to be indicative of a relapse of depressive illness, but without hospitalized. The onset of the event was used for the date of relapse.
Time Frame: Week 32
Population: The FAS includes all randomized participants.
Measure: Number; unit: Percentage of Participants
Arm/Group | Esketamine Nasal Spray + Oral Antidepressant (AD) | Quetiapine Extended Release (XR) + Oral AD
Number analyzed (Participants) | 336 | 340
Percentage of Participants | 21.7 | 14.1

3. Secondary Outcome: Change From Baseline in Clinician-rated Overall MADRS Score
Description: Change from baseline in clinician-rated overall MADRS score was reported. The MADRS is a clinician-rated scale designed to measure depression severity and to detect changes due to antidepressant treatment. The scale consists of 10 items, each of which is scored from 0 (item is not present or is normal) to 6 (severe or continuous presence of the symptoms), summed up for a total possible score range of 0 to 60. Higher scores represent a more severe condition. The MADRS evaluates apparent sadness, reported sadness, inner tension, sleep, appetite, concentration, lassitude, interest level, pessimistic thoughts, and suicidal thoughts.
Time Frame: Baseline, Weeks 1, 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 28, 30, 32
Population: The FAS included all randomized participants. Here, 'N' (number of participants analyzed) signifies participants evaluable for this outcome measure. Here, 'n' (number analyzed) signifies participants evaluable for this outcome measure at specified time points.
Measure: Mean (Standard Deviation); unit: Unit on scale
Arm/Group | Esketamine Nasal Spray + Oral Antidepressant (AD) | Quetiapine Extended Release (XR) + Oral AD
Number analyzed (Participants) | 327 | 330
Unit on scale
  Week 1: number analyzed (Participants) | 325 | 326
  Week 1 | -5.3 (5.71) | -3.7 (4.65)
  Week 2: number analyzed (Participants) | 324 | 315
  Week 2 | -9.0 (6.87) | -6.1 (6.52)
  Week 4: number analyzed (Participants) | 317 | 295
  Week 4 | -12.8 (7.50) | -9.8 (7.32)
  Week 6: number analyzed (Participants) | 312 | 285
  Week 6 | -14.9 (8.27) | -12.2 (8.11)
  Week 8: number analyzed (Participants) | 300 | 265
  Week 8 | -16.4 (8.67) | -14.3 (8.26)
  Week 10: number analyzed (Participants) | 288 | 242
  Week 10 | -18.2 (8.32) | -16.2 (7.38)
  Week 12: number analyzed (Participants) | 285 | 235
  Week 12 | -18.4 (8.26) | -16.7 (8.16)
  Week 14: number analyzed (Participants) | 280 | 232
  Week 14 | -19.0 (8.06) | -17.1 (8.06)
  Week 16: number analyzed (Participants) | 277 | 223
  Week 16 | -19.6 (8.16) | -17.8 (8.23)
  Week 18: number analyzed (Participants) | 267 | 219
  Week 18 | -19.9 (8.59) | -18.1 (8.36)
  Week 20: number analyzed (Participants) | 269 | 214
  Week 20 | -20.1 (8.75) | -19.1 (8.11)
  Week 22: number analyzed (Participants) | 263 | 214
  Week 22 | -20.6 (8.32) | -19.5 (8.04)
  Week 24: number analyzed (Participants) | 259 | 209
  Week 24 | -21.0 (8.58) | -20.1 (7.96)
  Week 26: number analyzed (Participants) | 257 | 206
  Week 26 | -21.2 (8.19) | -20.0 (8.18)
  Week 28: number analyzed (Participants) | 252 | 205
  Week 28 | -21.5 (8.33) | -20.8 (8.33)
  Week 30: number analyzed (Participants) | 250 | 200
  Week 30 | -21.8 (8.66) | -20.6 (8.39)
  Week 32: number analyzed (Participants) | 255 | 203
  Week 32 | -22.2 (8.12) | -20.5 (8.58)

4. Secondary Outcome: Change From Baseline in Clinician-rated Overall MADRS Score at Last Observation Carried Forward (LOCF)
Description: Change from baseline in clinician-rated overall MADRS score at LOCF was reported. The MADRS is a clinician-rated scale designed to measure depression severity and to detect changes due to antidepressant treatment. The scale consists of 10 items, each of which is scored from 0 (item is not present or is normal) to 6 (severe or continuous presence of the symptoms), summed up for a total possible score range of 0 to 60. Higher scores represent a more severe condition. The MADRS evaluates apparent sadness, reported sadness, inner tension, sleep, appetite, concentration, lassitude, interest level, pessimistic thoughts, and suicidal thoughts. LOCF is defined as the participants who had a missing value or who stopped treatment at a specific time point had their last non-missing value carried forward.
Time Frame: Baseline, LOCF at Weeks 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 28, 30, 32
Population: The FAS included all randomized participants. Here, 'N' (number of participants analyzed) signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Unit on scale
Arm/Group | Esketamine Nasal Spray + Oral Antidepressant (AD) | Quetiapine Extended Release (XR) + Oral AD
Number analyzed (Participants) | 327 | 330
Unit on scale
  Week 2 | -9.0 (6.86) | -5.8 (6.53)
  Week 4 | -12.6 (7.63) | -8.9 (7.70)
  Week 6 | -14.5 (8.47) | -10.7 (8.78)
  Week 8 | -15.7 (9.07) | -12.0 (9.30)
  Week 10 | -16.9 (9.15) | -12.8 (9.24)
  Week 12 | -17.1 (9.22) | -13.1 (9.82)
  Week 14 | -17.6 (9.08) | -13.2 (9.88)
  Week 16 | -18.1 (9.24) | -13.7 (10.17)
  Week 18 | -18.1 (9.60) | -13.8 (10.26)
  Week 20 | -18.2 (9.80) | -14.3 (10.46)
  Week 22 | -18.7 (9.83) | -14.6 (10.56)
  Week 24 | -18.8 (9.88) | -14.8 (10.77)
  Week 26 | -19.0 (9.76) | -14.9 (10.76)
  Week 28 | -19.1 (9.88) | -15.2 (11.08)
  Week 30 | -19.2 (10.10) | -15.2 (11.11)
  Week 32 | -19.6 (9.94) | -15.1 (11.18)

5. Secondary Outcome: Change From Baseline in Clinician-rated Overall Severity of Depressive Illness as Assessed by Clinical Global Impression - Severity (CGI-S) Scale Score
Description: Change from baseline in clinician-rated overall severity of depressive illness as assessed by CGI-S scale score was reported. The CGI-S provides an overall clinician-determined summary measure of the severity of the participant's illness that takes into account all available information, including knowledge of the participant's history, psychosocial circumstances, symptoms, behavior, and the impact of the symptoms on the participant's ability to function. The CGI-S evaluates the severity of psychopathology on a scale of 1 to 7. Considering total clinical experience, a participant is assessed on severity of mental illness at the time of rating according to: 1 = normal (not at all ill); 2 = borderline mentally ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; 7 = among the most extremely ill participants. Negative change in score indicates improvement.
Time Frame: Baseline, Weeks 1, 2, 3, 4, 8, 12, 16, 20, 24, 28, 32
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Esketamine Nasal Spray + Oral Antidepressant (AD) | Quetiapine Extended Release (XR) + Oral AD
Number analyzed (Participants) | 327 | 331
Units on scale
  Week 1: number analyzed (Participants) | 326 | 327
  Week 1 | -0.3 (0.58) | -0.2 (0.53)
  Week 2: number analyzed (Participants) | 324 | 314
  Week 2 | -0.7 (0.79) | -0.5 (0.77)
  Week 3: number analyzed (Participants) | 313 | 302
  Week 3 | -1.0 (0.88) | -0.7 (0.83)
  Week 4: number analyzed (Participants) | 317 | 296
  Week 4 | -1.3 (0.94) | -1.0 (0.95)
  Week 8: number analyzed (Participants) | 300 | 265
  Week 8 | -1.7 (0.98) | -1.4 (1.05)
  Week 12: number analyzed (Participants) | 286 | 238
  Week 12 | -1.9 (1.00) | -1.7 (1.07)
  Week 16: number analyzed (Participants) | 280 | 229
  Week 16 | -2.1 (1.05) | -1.9 (1.15)
  Week 20: number analyzed (Participants) | 270 | 218
  Week 20 | -2.2 (1.04) | -2.0 (1.22)
  Week 24: number analyzed (Participants) | 260 | 213
  Week 24 | -2.3 (1.06) | -2.1 (1.22)
  Week 28: number analyzed (Participants) | 255 | 208
  Week 28 | -2.4 (1.02) | -2.2 (1.19)
  Week 32: number analyzed (Participants) | 255 | 203
  Week 32 | -2.5 (1.05) | -2.3 (1.21)

6. Secondary Outcome: Change From Baseline in Clinician-rated Overall Severity of Depressive Illness as Assessed by CGI-S Scale Score at LOCF
Description: Change from Baseline in clinician-rated overall severity of depressive illness as assessed by CGI-S scale score at LOCF was reported. The CGI-S provides an overall clinician-determined summary measure of the severity of the participant's illness that takes into account all available information, including knowledge of the participant's history, psychosocial circumstances, symptoms, behavior, and the impact of the symptoms on the participant's ability to function. The CGI-S evaluates the severity of psychopathology on a scale of 1 to 7. A participant is assessed on severity of mental illness at the time of rating according to: 1 = normal (not at all ill); 2 = borderline mentally ill; 3 = mildly ill; 4 = moderately ill; 5 = markedly ill; 6 = severely ill; 7 = among the most extremely ill participants. LOCF is defined as the participants who had a missing value or who stopped treatment at a specific time point had their last non-missing value carried forward.
Time Frame: Baseline, LOCF at Weeks 2, 3, 4, 8, 12, 16, 20, 24, 28, 32
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Esketamine Nasal Spray + Oral Antidepressant (AD) | Quetiapine Extended Release (XR) + Oral AD
Number analyzed (Participants) | 327 | 331
Units on scale
  Week 2 | -0.7 (0.79) | -0.5 (0.75)
  Week 3 | -1.0 (0.88) | -0.7 (0.84)
  Week 4 | -1.3 (0.95) | -0.9 (0.96)
  Week 8 | -1.6 (1.02) | -1.2 (1.10)
  Week 12 | -1.8 (1.09) | -1.3 (1.18)
  Week 16 | -1.9 (1.16) | -1.4 (1.26)
  Week 20 | -2.0 (1.17) | -1.5 (1.32)
  Week 24 | -2.1 (1.22) | -1.5 (1.35)
  Week 28 | -2.1 (1.22) | -1.6 (1.36)
  Week 32 | -2.2 (1.27) | -1.6 (1.40)

7. Secondary Outcome: Clinician-rated Overall Severity of Depressive Illness as Assessed by Clinical Global Impression - Change (CGI-C) Scale Score
Description: Clinician-rated overall severity of depressive illness as assessed by CGI-C scale score was reported. The CGI-C evaluates the total improvement whether or not entirely due to drug treatment on a scale of 1 to 7. Compared to the condition at baseline, a participant is assessed on how much he/she has changed, according to: 1 = very much improved; 2 = much improved; 3 = minimally improved; 4 = no change; 5 = minimally worse; 6 = much worse; 7 = very much worse. Higher scores indicate more severity.
Time Frame: Baseline, Weeks 1, 2, 3, 4, 8, 12, 16, 20, 24, 28, 32
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Esketamine Nasal Spray + Oral Antidepressant (AD) | Quetiapine Extended Release (XR) + Oral AD
Number analyzed (Participants) | 327 | 331
Units on scale
  Week 1: number analyzed (Participants) | 326 | 327
  Week 1 | 3.3 (0.77) | 3.6 (0.72)
  Week 2: number analyzed (Participants) | 324 | 314
  Week 2 | 2.9 (0.87) | 3.3 (0.85)
  Week 3: number analyzed (Participants) | 313 | 302
  Week 3 | 2.7 (0.83) | 3.1 (0.84)
  Week 4: number analyzed (Participants) | 317 | 296
  Week 4 | 2.4 (0.85) | 2.9 (0.96)
  Week 8: number analyzed (Participants) | 300 | 265
  Week 8 | 2.1 (0.84) | 2.4 (0.93)
  Week 12: number analyzed (Participants) | 286 | 239
  Week 12 | 2.0 (0.85) | 2.3 (0.89)
  Week 16: number analyzed (Participants) | 280 | 229
  Week 16 | 1.9 (0.87) | 2.2 (0.99)
  Week 20: number analyzed (Participants) | 270 | 218
  Week 20 | 1.8 (0.85) | 2.1 (0.92)
  Week 24: number analyzed (Participants) | 260 | 213
  Week 24 | 1.8 (0.85) | 2.0 (0.84)
  Week 28: number analyzed (Participants) | 255 | 208
  Week 28 | 1.7 (0.84) | 2.0 (0.91)
  Week 32: number analyzed (Participants) | 255 | 203
  Week 32 | 1.6 (0.81) | 1.9 (0.88)

8. Secondary Outcome: Number of Participants With Clinician-rated Overall Severity of Depressive Illness as Assessed by CGI-C Scale Score at LOCF
Description: Number of participants with clinician-rated overall severity of depressive illness as assessed by CGI-C scale score at LOCF was reported. The CGI-C evaluates the total improvement whether or not entirely due to drug treatment on a scale of 1 to 7. Compared to the condition at baseline, a participant is assessed on how much he/she has changed, according to: 1 = very much improved; 2 = much improved; 3 = minimally improved; 4 = no change; 5 = minimally worse; 6 = much worse; 7 = very much worse. Higher scores indicate more severity. LOCF is defined as the participants who had a missing value or who stopped treatment at a specific time point had their last non-missing value carried forward.
Time Frame: Baseline, LOCF at Weeks 2, 3, 4, 8, 12, 16, 20, 24, 28, 32
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Esketamine Nasal Spray + Oral Antidepressant (AD) | Quetiapine Extended Release (XR) + Oral AD
Number analyzed (Participants) | 327 | 331
Participants
  Very much improved at Week 2 | 6 | 4
  Much improved at Week 2 | 97 | 39
  Minimally improved at Week 2 | 141 | 149
  No change at Week 2 | 75 | 108
  Minimally worse at Week 2 | 6 | 26
  Much worse at Week 2 | 1 | 5
  Very much worse at Week 2 | 1 | 0
  Very much improved at Week 3 | 14 | 8
  Much improved at Week 3 | 126 | 57
  Minimally improved at Week 3 | 135 | 159
  No change at Week 3 | 45 | 81
  Minimally worse at Week 3 | 6 | 20
  Much worse at Week 3 | 0 | 6
  Very much worse at Week 3 | 1 | 0
  Very much improved at Week 4 | 41 | 17
  Much improved at Week 4 | 150 | 83
  Minimally improved at Week 4 | 102 | 152
  No change at Week 4 | 29 | 52
  Minimally worse at Week 4 | 4 | 17
  Much worse at Week 4 | 0 | 10
  Very much worse at Week 4 | 1 | 0
  Very much improved at Week 8 | 68 | 38
  Much improved at Week 8 | 165 | 118
  Minimally improved at Week 8 | 68 | 105
  No change at Week 8 | 18 | 44
  Minimally worse at Week 8 | 5 | 16
  Much worse at Week 8 | 2 | 10
  Very much worse at Week 8 | 1 | 0
  Very much improved at Week 12 | 83 | 45
  Much improved at Week 12 | 156 | 120
  Minimally improved at Week 12 | 53 | 92
  No change at Week 12 | 24 | 47
  Minimally worse at Week 12 | 9 | 18
  Much worse at Week 12 | 1 | 9
  Very much worse at Week 12 | 1 | 0
  Very much improved at Week 16 | 100 | 55
  Much improved at Week 16 | 136 | 111
  Minimally improved at Week 16 | 58 | 84
  No change at Week 16 | 25 | 49
  Minimally worse at Week 16 | 5 | 23
  Much worse at Week 16 | 2 | 9
  Very much worse at Week 16 | 1 | 0
  Very much improved at Week 20 | 106 | 61
  Much improved at Week 20 | 137 | 110
  Minimally improved at Week 20 | 55 | 83
  No change at Week 20 | 19 | 49
  Minimally worse at Week 20 | 7 | 19
  Much worse at Week 20 | 2 | 9
  Very much worse at Week 20 | 1 | 0
  Very much improved at Week 24 | 123 | 64
  Much improved at Week 24 | 123 | 109
  Minimally improved at Week 24 | 48 | 86
  No change at Week 24 | 25 | 44
  Minimally worse at Week 24 | 6 | 19
  Much worse at Week 24 | 1 | 9
  Very much worse at Week 24 | 1 | 0
  Very much improved at Week 28 | 127 | 71
  Much improved at Week 28 | 121 | 104
  Minimally improved at Week 28 | 46 | 80
  No change at Week 28 | 24 | 48
  Minimally worse at Week 28 | 7 | 19
  Much worse at Week 28 | 1 | 9
  Very much worse at Week 28 | 1 | 0
  Very much improved at Week 32 | 148 | 82
  Much improved at Week 32 | 103 | 96
  Minimally improved at Week 32 | 42 | 81
  No change at Week 32 | 28 | 43
  Minimally worse at Week 32 | 4 | 20
  Much worse at Week 32 | 1 | 9
  Very much worse at Week 32 | 1 | 0

9. Secondary Outcome: Change From Baseline in Participant-reported Depressive Symptoms as Assessed by Patient Health Questionnaire (PHQ) 9-item Total Score
Description: Change from baseline in participant-reported depressive symptoms as assessed by PHQ 9-item total score was reported. The PHQ-9 is a validated 9-item, patient-reported outcome (PRO) measure to assess depressive symptoms. Each item is rated on a 4-point scale (0=not at all, 1=several days, 2=more than half the days, and 3=nearly every day). The participant's item responses are summed to provide a total score (range of 0 to 27), with higher scores indicating greater severity of depressive symptoms. The severity of the PHQ-9 is categorized as follows: None-minimal (0-4), Mild (5-9), Moderate (10-14), Moderately Severe (15-19) and Severe (20-27).
Time Frame: Baseline, Weeks 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 28, 30, 32
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Esketamine Nasal Spray + Oral Antidepressant (AD) | Quetiapine Extended Release (XR) + Oral AD
Number analyzed (Participants) | 322 | 316
Units on scale
  Week 2: number analyzed (Participants) | 319 | 310
  Week 2 | -4.9 (4.90) | -3.1 (4.62)
  Week 4: number analyzed (Participants) | 310 | 291
  Week 4 | -6.7 (5.25) | -5.0 (5.06)
  Week 6: number analyzed (Participants) | 305 | 278
  Week 6 | -8.1 (5.37) | -6.1 (5.64)
  Week 8: number analyzed (Participants) | 295 | 254
  Week 8 | -8.9 (5.74) | -7.4 (5.58)
  Week 10: number analyzed (Participants) | 282 | 236
  Week 10 | -9.6 (5.37) | -8.4 (5.58)
  Week 12: number analyzed (Participants) | 278 | 227
  Week 12 | -9.8 (5.78) | -8.7 (5.65)
  Week 14: number analyzed (Participants) | 273 | 224
  Week 14 | -10.2 (5.49) | -8.5 (5.76)
  Week 16: number analyzed (Participants) | 274 | 216
  Week 16 | -10.5 (5.50) | -9.2 (5.77)
  Week 18: number analyzed (Participants) | 260 | 212
  Week 18 | -10.6 (5.79) | -9.3 (5.74)
  Week 20: number analyzed (Participants) | 264 | 209
  Week 20 | -10.4 (5.64) | -9.4 (5.97)
  Week 22: number analyzed (Participants) | 261 | 209
  Week 22 | -10.7 (5.74) | -9.5 (5.87)
  Week 24: number analyzed (Participants) | 257 | 206
  Week 24 | -10.6 (5.84) | -9.7 (6.08)
  Week 26: number analyzed (Participants) | 255 | 201
  Week 26 | -10.9 (5.88) | -9.7 (6.21)
  Week 28: number analyzed (Participants) | 250 | 201
  Week 28 | -10.9 (6.16) | -10.0 (6.23)
  Week 30: number analyzed (Participants) | 248 | 197
  Week 30 | -11.2 (6.39) | -10.1 (6.08)
  Week 32: number analyzed (Participants) | 253 | 198
  Week 32 | -11.4 (6.40) | -10.5 (6.01)

10. Secondary Outcome: Change From Baseline in Participant-reported Depressive Symptoms as Assessed by PHQ 9-item Total Score at LOCF
Description: Change from baseline in participant-reported depressive symptoms as assessed by PHQ 9-item total score at LOCF was reported. The PHQ-9 is a validated 9-item, PRO measure to assess depressive symptoms. Each item is rated on a 4-point scale (0=not at all, 1=several days, 2=more than half the days, and 3=nearly every day). The participant's item responses are summed to provide a total score (range of 0 to 27), with higher scores indicating greater severity of depressive symptoms. The severity of the PHQ-9 is categorized as follows: None-minimal (0-4), Mild (5-9), Moderate (10-14), Moderately Severe (15-19) and Severe (20-27). LOCF is defined as participants who had a missing value or who stopped treatment at a specific time point had their last non-missing value carried forward.
Time Frame: Baseline, LOCF at Weeks 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 22, 24, 26, 28, 30, 32
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Esketamine Nasal Spray + Oral Antidepressant (AD) | Quetiapine Extended Release (XR) + Oral AD
Number analyzed (Participants) | 322 | 316
Units on scale
  Week 2: number analyzed (Participants) | 319 | 310
  Week 2 | -4.9 (4.90) | -3.1 (4.62)
  Week 4: number analyzed (Participants) | 320 | 314
  Week 4 | -6.6 (5.33) | -4.7 (5.06)
  Week 6: number analyzed (Participants) | 320 | 315
  Week 6 | -7.8 (5.51) | -5.6 (5.69)
  Week 8: number analyzed (Participants) | 322 | 315
  Week 8 | -8.5 (5.94) | -6.3 (5.86)
  Week 10 | -9.0 (5.75) | -7.0 (5.90)
  Week 12 | -9.1 (6.13) | -7.1 (6.07)
  Week 14 | -9.3 (5.93) | -6.9 (6.12)
  Week 16 | -9.6 (5.98) | -7.4 (6.20)
  Week 18 | -9.5 (6.26) | -7.3 (6.21)
  Week 20 | -9.4 (6.12) | -7.4 (6.32)
  Week 22 | -9.7 (6.27) | -7.5 (6.31)
  Week 24 | -9.5 (6.35) | -7.5 (6.47)
  Week 26 | -9.7 (6.46) | -7.5 (6.56)
  Week 28 | -9.7 (6.66) | -7.6 (6.64)
  Week 30 | -9.9 (6.85) | -7.6 (6.61)
  Week 32 | -10.1 (6.94) | -8.0 (6.70)

11. Secondary Outcome: Change From Baseline in Participant-reported Functional Impairment and Associated Disability as Assessed by Sheehan Disability Scale (SDS) Total Score
Description: Change from baseline in participant-reported functional impairment and associated disability as assessed by SDS total score was reported. The SDS is a validated PRO measure consisting of a 5-item questionnaire that has been widely used and accepted for assessment of functional impairment and associated disability. The first 3 items assess disruption of (1) work/school, (2) social life, and (3) family life/home responsibilities using a rating scale from 0 to 10. It also has 1 item assessing days lost from school or work and 1 item assessing days of underproductivity. The scores for the first 3 items are summed to create a total score of 0 to 30, where higher score indicates greater impairment. Scores <=2 for each item and <= 6 for the total score are considered functional remission.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Esketamine Nasal Spray + Oral Antidepressant (AD) | Quetiapine Extended Release (XR) + Oral AD
Number analyzed (Participants) | 310 | 303
Units on scale
  Week 4: number analyzed (Participants) | 307 | 298
  Week 4 | -5.9 (6.58) | -4.1 (5.89)
  Week 8: number analyzed (Participants) | 284 | 252
  Week 8 | -8.6 (7.03) | -6.8 (7.63)
  Week 12: number analyzed (Participants) | 272 | 232
  Week 12 | -9.7 (7.54) | -8.6 (6.94)
  Week 16: number analyzed (Participants) | 268 | 219
  Week 16 | -10.6 (7.29) | -9.0 (7.50)
  Week 20: number analyzed (Participants) | 258 | 208
  Week 20 | -10.9 (7.57) | -9.0 (7.41)
  Week 24: number analyzed (Participants) | 249 | 201
  Week 24 | -11.2 (7.88) | -10.1 (7.76)
  Week 28: number analyzed (Participants) | 245 | 200
  Week 28 | -11.9 (7.84) | -10.8 (8.03)
  Week 32: number analyzed (Participants) | 244 | 193
  Week 32 | -12.6 (8.09) | -11.1 (8.06)

12. Secondary Outcome: Change From Baseline in Participant-reported Functional Impairment and Associated Disability as Assessed by SDS Total Score at LOCF
Description: Change from baseline in participant-reported functional impairment and associated disability as assessed by SDS total score at LOCF was reported. The SDS is a validated PRO measure consisting of a 5-item questionnaire for assessment of functional impairment and associated disability. The first 3 items assess disruption of (1) work/school, (2) social life, and (3) family life/home responsibilities using a rating scale from 0 to 10. It also has 1 item assessing days lost from school or work and 1 item assessing days of underproductivity. The scores for the first 3 items are summed to create a total score of 0 to 30, where higher score indicates greater impairment. Scores <=2 for each item and <= 6 for the total score are considered functional remission. LOCF is defined as the participants who had a missing value or who stopped treatment at a specific time point had their last non-missing value carried forward.
Time Frame: Baseline, LOCF at Weeks 4, 8, 12, 16, 20, 24, 28, 32
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Esketamine Nasal Spray + Oral Antidepressant (AD) | Quetiapine Extended Release (XR) + Oral AD
Number analyzed (Participants) | 310 | 303
Units on scale
  Week 4: number analyzed (Participants) | 307 | 298
  Week 4 | -5.9 (6.58) | -4.1 (5.89)
  Week 8: number analyzed (Participants) | 309 | 303
  Week 8 | -8.2 (7.06) | -5.8 (7.45)
  Week 12 | -9.0 (7.59) | -6.8 (7.59)
  Week 16 | -9.8 (7.47) | -7.0 (7.99)
  Week 20 | -9.9 (7.75) | -7.0 (7.97)
  Week 24 | -10.0 (8.13) | -7.6 (8.37)
  Week 28 | -10.4 (8.21) | -7.9 (8.69)
  Week 32 | -11.1 (8.56) | -8.2 (8.78)

13. Secondary Outcome: Change From Baseline in Participant-reported Health-related Quality of Life (HRQoL) and Health Status as Assessed by 36-item Short-Form Health Survey (SF-36) Scale Score
Description: Change from baseline in participant-reported HRQoL and health status as assessed by SF-36 scale score was reported. The SF-36 consists of 8 subscales (physical function, role limitations due to physical problems, pain, general health perception, vitality, social function, role limitations due to emotional problems, and mental health). Participants self-report on items in a subscale that have between 2-6 choices per item using likert-type responses (for example: none of the time, some of the time, etc.). Summations of item scores of the same subscale give the subscale scores, which are transformed into a range from 0 to 100; 0= worst HRQoL, 100=best HRQoL. Higher scores indicate better health status.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32
Population: The FAS included all randomized participants. Here, 'N' (number of participants analyzed) signifies participants evaluable for this outcome measure. Here, 'n' (number analyzed) signifies participants evaluable for this outcome measure at specified categories with time points.
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Esketamine Nasal Spray + Oral Antidepressant (AD) | Quetiapine Extended Release (XR) + Oral AD
Number analyzed (Participants) | 319 | 308
Units on scale
  Physical Functioning Week 4: number analyzed (Participants) | 310 | 295
  Physical Functioning Week 4 | 3.5 (7.16) | 2.2 (6.85)
  Physical Functioning Week 8: number analyzed (Participants) | 287 | 250
  Physical Functioning Week 8 | 5.4 (7.64) | 3.8 (8.19)
  Physical Functioning Week 12: number analyzed (Participants) | 274 | 228
  Physical Functioning Week 12 | 5.8 (8.29) | 4.7 (8.00)
  Physical Functioning Week 16: number analyzed (Participants) | 268 | 216
  Physical Functioning Week 16 | 6.2 (8.36) | 5.2 (8.42)
  Physical Functioning Week 20: number analyzed (Participants) | 258 | 207
  Physical Functioning Week 20 | 6.1 (8.62) | 5.1 (8.87)
  Physical Functioning Week 24: number analyzed (Participants) | 252 | 197
  Physical Functioning Week 24 | 6.2 (9.01) | 5.9 (9.23)
  Physical Functioning Week 28: number analyzed (Participants) | 246 | 197
  Physical Functioning Week 28 | 6.4 (8.68) | 6.2 (9.51)
  Physical Functioning Week 32: number analyzed (Participants) | 250 | 195
  Physical Functioning Week 32 | 6.8 (8.79) | 6.4 (9.58)
  Role-Physical Week 4: number analyzed (Participants) | 314 | 299
  Role-Physical Week 4 | 5.7 (9.57) | 3.1 (9.75)
  Role-Physical Week 8: number analyzed (Participants) | 291 | 251
  Role-Physical Week 8 | 7.5 (10.49) | 6.1 (11.67)
  Role-Physical Week 12: number analyzed (Participants) | 276 | 229
  Role-Physical Week 12 | 8.8 (10.59) | 7.1 (11.38)
  Role-Physical Week 16: number analyzed (Participants) | 272 | 218
  Role-Physical Week 16 | 10.0 (11.60) | 8.3 (12.47)
  Role-Physical Week 20: number analyzed (Participants) | 264 | 206
  Role-Physical Week 20 | 10.0 (11.75) | 8.2 (12.34)
  Role-Physical Week 24: number analyzed (Participants) | 256 | 203
  Role-Physical Week 24 | 10.4 (11.97) | 9.2 (12.50)
  Role-Physical Week 28: number analyzed (Participants) | 250 | 199
  Role-Physical Week 28 | 10.9 (11.92) | 8.8 (12.62)
  Role-Physical Week 32: number analyzed (Participants) | 250 | 196
  Role-Physical Week 32 | 11.7 (11.97) | 9.4 (12.39)
  Body Pain Week 4: number analyzed (Participants) | 315 | 308
  Body Pain Week 4 | 3.7 (9.05) | 2.3 (8.50)
  Body Pain Week 8: number analyzed (Participants) | 294 | 254
  Body Pain Week 8 | 4.5 (10.04) | 4.0 (8.85)
  Body Pain Week 12: number analyzed (Participants) | 280 | 235
  Body Pain Week 12 | 5.1 (9.93) | 5.3 (9.71)
  Body Pain Week 16: number analyzed (Participants) | 275 | 224
  Body Pain Week 16 | 5.6 (10.05) | 5.5 (10.52)
  Body Pain Week 20: number analyzed (Participants) | 265 | 215
  Body Pain Week 20 | 5.7 (11.14) | 6.0 (10.41)
  Body Pain Week 24: number analyzed (Participants) | 255 | 209
  Body Pain Week 24 | 6.2 (10.68) | 6.1 (10.64)
  Body Pain Week 28: number analyzed (Participants) | 251 | 204
  Body Pain Week 28 | 6.2 (11.32) | 6.3 (11.34)
  Body Pain Week 32: number analyzed (Participants) | 252 | 201
  Body Pain Week 32 | 6.7 (11.03) | 7.2 (11.62)
  General Health Week 4: number analyzed (Participants) | 315 | 302
  General Health Week 4 | 5.3 (7.85) | 3.3 (7.45)
  General Health Week 8: number analyzed (Participants) | 289 | 252
  General Health Week 8 | 7.2 (8.63) | 5.7 (8.50)
  General Health Week 12: number analyzed (Participants) | 278 | 232
  General Health Week 12 | 7.9 (8.79) | 6.4 (9.02)
  General Health Week 16: number analyzed (Participants) | 274 | 221
  General Health Week 16 | 8.8 (9.09) | 7.3 (9.55)
  General Health Week 20: number analyzed (Participants) | 267 | 212
  General Health Week 20 | 9.0 (9.30) | 7.2 (9.71)
  General Health Week 24: number analyzed (Participants) | 255 | 207
  General Health Week 24 | 9.5 (9.73) | 7.7 (10.05)
  General Health Week 28: number analyzed (Participants) | 249 | 200
  General Health Week 28 | 10.1 (9.71) | 8.8 (10.38)
  General Health Week 32: number analyzed (Participants) | 253 | 198
  General Health Week 32 | 10.6 (10.25) | 9.7 (10.33)
  Vitality Week 4: number analyzed (Participants) | 319 | 301
  Vitality Week 4 | 8.7 (9.13) | 5.2 (7.75)
  Vitality Week 8: number analyzed (Participants) | 293 | 249
  Vitality Week 8 | 11.3 (10.04) | 9.2 (9.44)
  Vitality Week 12: number analyzed (Participants) | 277 | 230
  Vitality Week 12 | 12.4 (10.36) | 10.8 (9.79)
  Vitality Week 16: number analyzed (Participants) | 276 | 220
  Vitality Week 16 | 13.1 (10.69) | 12.1 (9.88)
  Vitality Week 20: number analyzed (Participants) | 267 | 210
  Vitality Week 20 | 13.2 (10.67) | 12.6 (10.64)
  Vitality Week 24: number analyzed (Participants) | 251 | 206
  Vitality Week 24 | 13.4 (10.83) | 12.9 (11.26)
  Vitality Week 28: number analyzed (Participants) | 251 | 203
  Vitality Week 28 | 14.2 (11.25) | 13.9 (11.19)
  Vitality Week 32: number analyzed (Participants) | 251 | 198
  Vitality Week 32 | 15.2 (11.64) | 14.0 (11.34)
  Social Functioning Week 4: number analyzed (Participants) | 304 | 300
  Social Functioning Week 4 | 7.1 (10.32) | 5.0 (8.83)
  Social Functioning Week 8: number analyzed (Participants) | 284 | 251
  Social Functioning Week 8 | 11.2 (11.42) | 8.7 (9.59)
  Social Functioning Week 12: number analyzed (Participants) | 274 | 231
  Social Functioning Week 12 | 12.4 (11.29) | 10.2 (10.45)
  Social Functioning Week 16: number analyzed (Participants) | 269 | 220
  Social Functioning Week 16 | 13.5 (10.92) | 11.2 (11.24)
  Social Functioning Week 20: number analyzed (Participants) | 258 | 208
  Social Functioning Week 20 | 13.6 (11.65) | 11.7 (10.73)
  Social Functioning Week 24: number analyzed (Participants) | 247 | 206
  Social Functioning Week 24 | 14.3 (11.55) | 12.5 (11.75)
  Social Functioning Week 28: number analyzed (Participants) | 241 | 198
  Social Functioning Week 28 | 15.3 (11.26) | 13.3 (11.15)
  Social Functioning Week 32: number analyzed (Participants) | 245 | 197
  Social Functioning Week 32 | 16.1 (11.34) | 13.8 (11.47)
  Role-Emotional Week 4: number analyzed (Participants) | 316 | 305
  Role-Emotional Week 4 | 8.6 (9.62) | 5.3 (9.53)
  Role-Emotional Week 8: number analyzed (Participants) | 293 | 254
  Role-Emotional Week 8 | 12.7 (10.67) | 10.1 (11.30)
  Role-Emotional Week 12: number analyzed (Participants) | 280 | 235
  Role-Emotional Week 12 | 13.8 (10.70) | 12.2 (11.48)
  Role-Emotional Week 16: number analyzed (Participants) | 277 | 224
  Role-Emotional Week 16 | 15.4 (11.30) | 13.2 (12.07)
  Role-Emotional Week 20: number analyzed (Participants) | 268 | 213
  Role-Emotional Week 20 | 15.8 (11.26) | 13.4 (11.14)
  Role-Emotional Week 24: number analyzed (Participants) | 257 | 209
  Role-Emotional Week 24 | 16.0 (11.79) | 14.7 (11.71)
  Role-Emotional Week 28: number analyzed (Participants) | 252 | 204
  Role-Emotional Week 28 | 17.3 (12.44) | 15.0 (11.58)
  Role-Emotional Week 32: number analyzed (Participants) | 252 | 201
  Role-Emotional Week 32 | 18.1 (12.49) | 14.9 (12.62)
  Mental Health Week 4: number analyzed (Participants) | 311 | 297
  Mental Health Week 4 | 9.8 (9.77) | 6.7 (9.34)
  Mental Health Week 8: number analyzed (Participants) | 287 | 248
  Mental Health Week 8 | 13.5 (10.37) | 11.6 (10.78)
  Mental Health Week 12: number analyzed (Participants) | 278 | 231
  Mental Health Week 12 | 15.0 (10.50) | 13.3 (10.84)
  Mental Health Week 16: number analyzed (Participants) | 267 | 217
  Mental Health Week 16 | 16.1 (11.04) | 14.3 (11.01)
  Mental Health Week 20: number analyzed (Participants) | 266 | 209
  Mental Health Week 20 | 16.5 (10.90) | 14.7 (11.36)
  Mental Health Week 24: number analyzed (Participants) | 251 | 204
  Mental Health Week 24 | 16.6 (11.69) | 15.3 (11.45)
  Mental Health Week 28: number analyzed (Participants) | 246 | 200
  Mental Health Week 28 | 17.6 (11.40) | 16.5 (12.16)
  Mental Health Week 32: number analyzed (Participants) | 251 | 195
  Mental Health Week 32 | 18.4 (11.89) | 17.0 (12.05)

14. Secondary Outcome: Change From Baseline in Participant-reported HRQoL and Health Status as Assessed by SF-36 Scale Score at LOCF
Description: Change from baseline in participant-reported HRQoL and health status as assessed by SF-36 domain scores at LOCF was reported. The SF-36 consists of 8 subscales (physical function, role limitations due to physical problems, pain, general health perception, vitality, social function, role limitations due to emotional problems, and mental health). Participants self-report on items in a subscale that have between 2-6 choices per item using likert-type responses (for example: none of the time, some of the time, etc.). Summations of item scores of the same subscale give the subscale scores, which are transformed into a range from 0 to 100; 0= worst HRQoL, 100=best HRQoL. Higher scores indicate better health status. LOCF is defined as participants who had a missing value or who stopped treatment at a specific time point had their last non-missing value carried forward.
Time Frame: Baseline, LOCF at Weeks 8, 12, 16, 20, 24, 28, 32
Population: The FAS included all randomized participants. Here, 'N' (number of participants analyzed) signifies participants evaluable for this outcome measure. Here, 'n' (number analyzed) signifies participants evaluable for this outcome measure at specified categories with time points. LOCF was applied only for participants whose questionnaire was completely missing. No LOCF imputation was done on partially completed questionnaire.
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Esketamine Nasal Spray + Oral Antidepressant (AD) | Quetiapine Extended Release (XR) + Oral AD
Number analyzed (Participants) | 319 | 308
Units on scale
  Physical Functioning Week 8: number analyzed (Participants) | 308 | 300
  Physical Functioning Week 8 | 5.1 (7.61) | 3.2 (8.15)
  Physical Functioning Week 12: number analyzed (Participants) | 308 | 299
  Physical Functioning Week 12 | 5.3 (8.22) | 3.9 (7.96)
  Physical Functioning Week 16: number analyzed (Participants) | 307 | 298
  Physical Functioning Week 16 | 5.6 (8.33) | 4.2 (8.27)
  Physical Functioning Week 20: number analyzed (Participants) | 306 | 300
  Physical Functioning Week 20 | 5.5 (8.63) | 4.0 (8.48)
  Physical Functioning Week 24: number analyzed (Participants) | 309 | 295
  Physical Functioning Week 24 | 5.6 (8.83) | 4.4 (8.84)
  Physical Functioning Week 28: number analyzed (Participants) | 309 | 298
  Physical Functioning Week 28 | 5.6 (8.71) | 4.5 (8.97)
  Physical Functioning Week 32: number analyzed (Participants) | 312 | 300
  Physical Functioning Week 32 | 6.0 (8.77) | 4.6 (9.05)
  Role-Physical Week 8: number analyzed (Participants) | 315 | 302
  Role-Physical Week 8 | 7.4 (10.51) | 5.3 (11.50)
  Role-Physical Week 12: number analyzed (Participants) | 313 | 301
  Role-Physical Week 12 | 8.3 (10.87) | 5.7 (11.31)
  Role-Physical Week 16: number analyzed (Participants) | 313 | 302
  Role-Physical Week 16 | 9.3 (11.49) | 6.2 (12.23)
  Role-Physical Week 20: number analyzed (Participants) | 314 | 298
  Role-Physical Week 20 | 9.1 (11.69) | 6.3 (12.09)
  Role-Physical Week 24: number analyzed (Participants) | 316 | 301
  Role-Physical Week 24 | 9.2 (11.93) | 6.9 (12.48)
  Role-Physical Week 28: number analyzed (Participants) | 316 | 301
  Role-Physical Week 28 | 9.4 (12.00) | 6.8 (12.36)
  Role-Physical Week 32: number analyzed (Participants) | 315 | 303
  Role-Physical Week 32 | 10.2 (12.21) | 7.2 (12.29)
  Body Pain Week 8: number analyzed (Participants) | 318 | 306
  Body Pain Week 8 | 4.4 (9.84) | 3.5 (8.79)
  Body Pain Week 12: number analyzed (Participants) | 317 | 307
  Body Pain Week 12 | 4.8 (9.99) | 4.2 (9.51)
  Body Pain Week 16: number analyzed (Participants) | 317 | 308
  Body Pain Week 16 | 5.2 (10.14) | 4.3 (10.02)
  Body Pain Week 20: number analyzed (Participants) | 316 | 308
  Body Pain Week 20 | 5.2 (10.85) | 4.5 (10.05)
  Body Pain Week 24: number analyzed (Participants) | 316 | 307
  Body Pain Week 24 | 5.6 (10.45) | 4.4 (10.26)
  Body Pain Week 28: number analyzed (Participants) | 318 | 307
  Body Pain Week 28 | 5.4 (11.01) | 4.5 (10.78)
  Body Pain Week 32: number analyzed (Participants) | 318 | 308
  Body Pain Week 32 | 6.0 (10.93) | 5.0 (11.10)
  General Health Week 8: number analyzed (Participants) | 313 | 303
  General Health Week 8 | 6.9 (8.85) | 4.9 (8.19)
  General Health Week 12: number analyzed (Participants) | 315 | 304
  General Health Week 12 | 7.4 (9.19) | 5.1 (8.68)
  General Health Week 16: number analyzed (Participants) | 316 | 305
  General Health Week 16 | 8.0 (9.41) | 5.6 (9.20)
  General Health Week 20: number analyzed (Participants) | 318 | 306
  General Health Week 20 | 8.1 (9.60) | 5.5 (9.37)
  General Health Week 24: number analyzed (Participants) | 316 | 306
  General Health Week 24 | 8.2 (10.08) | 5.6 (9.57)
  General Health Week 28: number analyzed (Participants) | 316 | 304
  General Health Week 28 | 8.6 (10.19) | 6.1 (10.01)
  General Health Week 32: number analyzed (Participants) | 319 | 306
  General Health Week 32 | 9.2 (10.78) | 6.7 (10.18)
  Vitality Week 8: number analyzed (Participants) | 317 | 299
  Vitality Week 8 | 11.1 (10.08) | 7.8 (9.46)
  Vitality Week 12: number analyzed (Participants) | 314 | 301
  Vitality Week 12 | 11.7 (10.48) | 8.7 (9.98)
  Vitality Week 16: number analyzed (Participants) | 317 | 303
  Vitality Week 16 | 12.3 (10.81) | 9.5 (10.26)
  Vitality Week 20: number analyzed (Participants) | 317 | 301
  Vitality Week 20 | 12.3 (10.94) | 9.6 (10.77)
  Vitality Week 24: number analyzed (Participants) | 311 | 303
  Vitality Week 24 | 12.2 (11.04) | 9.6 (11.34)
  Vitality Week 28: number analyzed (Participants) | 316 | 305
  Vitality Week 28 | 12.8 (11.43) | 10.1 (11.53)
  Vitality Week 32: number analyzed (Participants) | 315 | 304
  Vitality Week 32 | 13.8 (11.99) | 10.4 (11.65)
  Social Functioning Week 8: number analyzed (Participants) | 308 | 303
  Social Functioning Week 8 | 10.7 (11.31) | 7.6 (9.72)
  Social Functioning Week 12: number analyzed (Participants) | 310 | 301
  Social Functioning Week 12 | 11.4 (11.29) | 8.6 (10.47)
  Social Functioning Week 16: number analyzed (Participants) | 310 | 302
  Social Functioning Week 16 | 12.2 (11.24) | 9.0 (11.22)
  Social Functioning Week 20: number analyzed (Participants) | 307 | 299
  Social Functioning Week 20 | 12.3 (11.91) | 9.1 (10.92)
  Social Functioning Week 24: number analyzed (Participants) | 306 | 302
  Social Functioning Week 24 | 12.7 (11.81) | 9.5 (11.63)
  Social Functioning Week 28: number analyzed (Participants) | 306 | 299
  Social Functioning Week 28 | 13.0 (12.09) | 9.8 (11.49)
  Social Functioning Week 32: number analyzed (Participants) | 309 | 302
  Social Functioning Week 32 | 14.0 (12.35) | 10.3 (11.71)
  Role-Emotional Week 8: number analyzed (Participants) | 315 | 304
  Role-Emotional Week 8 | 12.0 (10.75) | 8.6 (11.30)
  Role-Emotional Week 12: number analyzed (Participants) | 315 | 306
  Role-Emotional Week 12 | 12.7 (10.89) | 9.8 (11.82)
  Role-Emotional Week 16: number analyzed (Participants) | 317 | 307
  Role-Emotional Week 16 | 14.2 (11.53) | 10.3 (12.32)
  Role-Emotional Week 20: number analyzed (Participants) | 317 | 305
  Role-Emotional Week 20 | 14.3 (11.77) | 10.4 (11.67)
  Role-Emotional Week 24: number analyzed (Participants) | 316 | 306
  Role-Emotional Week 24 | 14.3 (12.15) | 11.2 (12.22)
  Role-Emotional Week 28: number analyzed (Participants) | 317 | 306
  Role-Emotional Week 28 | 15.2 (12.91) | 11.2 (12.30)
  Role-Emotional Week 32: number analyzed (Participants) | 316 | 307
  Role-Emotional Week 32 | 16.0 (13.16) | 11.2 (12.96)
  Mental Health Week 8: number analyzed (Participants) | 310 | 298
  Mental Health Week 8 | 12.9 (10.76) | 9.8 (11.04)
  Mental Health Week 12: number analyzed (Participants) | 313 | 301
  Mental Health Week 12 | 14.0 (11.09) | 10.6 (11.44)
  Mental Health Week 16: number analyzed (Participants) | 306 | 298
  Mental Health Week 16 | 14.7 (11.63) | 10.9 (11.85)
  Mental Health Week 20: number analyzed (Participants) | 313 | 299
  Mental Health Week 20 | 15.0 (11.64) | 11.2 (12.07)
  Mental Health Week 24: number analyzed (Participants) | 308 | 299
  Mental Health Week 24 | 14.8 (12.24) | 11.5 (12.23)
  Mental Health Week 28: number analyzed (Participants) | 308 | 300
  Mental Health Week 28 | 15.5 (12.35) | 12.2 (13.01)
  Mental Health Week 32: number analyzed (Participants) | 312 | 299
  Mental Health Week 32 | 16.3 (12.90) | 12.6 (13.08)

15. Secondary Outcome: Change From Baseline in Participant-reported Quality of Life as Assessed by Quality of Life in Depression Scale (QLDS) Total Score
Description: Change from baseline in participant-reported quality of life as assessed by QLDS total score was reported. The QLDS is a disease-specific validated PRO measure which assesses the impact that depression has on a participant's quality of life. It is a 34-item self-rated questionnaire which consists of dichotomous response questions, with the response being either True/Not True. Each statement on the QLDS is given a score of "1" or "0". A score of "1" is indicative of adverse quality of life. All item scores are summed to give a total score that ranges from 0 (good quality of life) to 34 (very poor quality of life). A higher score indicates a more severe condition.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on Scale
Arm/Group | Esketamine Nasal Spray + Oral Antidepressant (AD) | Quetiapine Extended Release (XR) + Oral AD
Number analyzed (Participants) | 318 | 305
Units on Scale
  Week 4: number analyzed (Participants) | 315 | 300
  Week 4 | -8.9 (8.83) | -5.6 (7.43)
  Week 8: number analyzed (Participants) | 292 | 253
  Week 8 | -12.0 (9.36) | -9.1 (9.31)
  Week 12: number analyzed (Participants) | 281 | 234
  Week 12 | -13.5 (9.30) | -10.9 (9.52)
  Week 16: number analyzed (Participants) | 277 | 221
  Week 16 | -14.2 (9.39) | -11.6 (9.39)
  Week 20: number analyzed (Participants) | 264 | 212
  Week 20 | -14.3 (9.50) | -12.1 (9.74)
  Week 24: number analyzed (Participants) | 256 | 205
  Week 24 | -14.9 (9.44) | -12.8 (9.64)
  Week 28: number analyzed (Participants) | 249 | 201
  Week 28 | -15.6 (9.42) | -13.7 (9.51)
  Week 32: number analyzed (Participants) | 252 | 198
  Week 32 | -16.0 (9.55) | -14.2 (9.96)

16. Secondary Outcome: Change From Baseline in Participant-reported Quality of Life as Assessed by QLDS Total Score at LOCF
Description: Change from baseline in participant-reported quality of life as assessed by QLDS total score at LOCF was reported. The QLDS is a disease-specific validated PRO measure which assesses the impact that depression has on a participant's quality of life. It is a 34-item self-rated questionnaire which consists of dichotomous response questions, with the response being either True/Not True. Each statement on the QLDS is given a score of "1" or "0". A score of "1" is indicative of adverse quality of life. All item scores are summed to give a total score that ranges from 0 (good quality of life) to 34 (very poor quality of life). A higher score indicates a more severe condition. LOCF is defined as the participants who had a missing value or who stopped treatment at a specific time point had their last non-missing value carried forward.
Time Frame: Baseline, LOCF at Weeks 4, 8, 12, 16, 20, 24, 28, 32
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on Scale
Arm/Group | Esketamine Nasal Spray + Oral Antidepressant (AD) | Quetiapine Extended Release (XR) + Oral AD
Number analyzed (Participants) | 318 | 305
Units on Scale
  Week 4: number analyzed (Participants) | 315 | 300
  Week 4 | -8.9 (8.83) | -5.6 (7.43)
  Week 8 | -11.3 (9.59) | -8.1 (9.22)
  Week 12 | -12.3 (9.73) | -9.0 (9.62)
  Week 16 | -13.0 (9.86) | -9.3 (9.80)
  Week 20 | -13.0 (9.93) | -9.5 (10.02)
  Week 24 | -13.3 (9.98) | -9.8 (10.18)
  Week 28 | -13.6 (10.06) | -10.3 (10.26)
  Week 32 | -14.1 (10.29) | -10.5 (10.59)

17. Secondary Outcome: Change From Baseline in Participant-reported Health-related Quality of Life as Assessed by EuroQol-5 Dimension-5 Level (EQ-5D-5L) Score: Health Status Index
Description: Change from baseline in participant-reported health-related quality of Life as assessed by EQ-5D-5L score: health status index was reported. The EQ-5D-5L is a standardized 2-part instrument used to measure health outcomes, primarily designed for self-completion by respondents. It consists of the EQ-5D-5L descriptive system and the EQ Visual Analogue Scale (EQ-VAS). The EQ-5D-5L descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each of the 5 dimensions is divided into 5 levels of perceived problems (level 1 = no problem, level 2 = slight problems, level 3 = moderate problems, level 4 = severe problems, level 5 = extreme problems). The participant selects an answer for each of the 5 dimensions considering the response that best matches his or her health "today." Responses were used to generate health status index which ranges from 0 (dead) and 1 (full health), a lower score indicates worse health.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on Scale
Arm/Group | Esketamine Nasal Spray + Oral Antidepressant (AD) | Quetiapine Extended Release (XR) + Oral AD
Number analyzed (Participants) | 320 | 308
Units on Scale
  Week 4: number analyzed (Participants) | 318 | 306
  Week 4 | 0.177 (0.2354) | 0.124 (0.2280)
  Week 8: number analyzed (Participants) | 296 | 258
  Week 8 | 0.234 (0.2655) | 0.206 (0.2463)
  Week 12: number analyzed (Participants) | 282 | 237
  Week 12 | 0.276 (0.2405) | 0.227 (0.2367)
  Week 16: number analyzed (Participants) | 277 | 225
  Week 16 | 0.284 (0.2445) | 0.232 (0.2431)
  Week 20: number analyzed (Participants) | 268 | 214
  Week 20 | 0.294 (0.2399) | 0.238 (0.2423)
  Week 24: number analyzed (Participants) | 258 | 209
  Week 24 | 0.297 (0.2498) | 0.259 (0.2489)
  Week 28: number analyzed (Participants) | 250 | 205
  Week 28 | 0.303 (0.2584) | 0.262 (0.2492)
  Week 32: number analyzed (Participants) | 254 | 200
  Week 32 | 0.317 (0.2636) | 0.279 (0.2581)

18. Secondary Outcome: Change From Baseline in Participant-reported Health-related Quality of Life Group, as Assessed by EQ-5D-5L Score: Health Status Index at LOCF
Description: Change from baseline in participant-reported health-related quality of Life as assessed by EQ-5D-5L score: health status index at LOCF was reported. The EQ-5D-5L is a standardized 2-part instrument used to measure health outcomes, primarily designed for self-completion by respondents. It consists of the EQ-5D-5L descriptive system and the EQ-VAS. The EQ-5D-5L descriptive system comprises of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each of the 5 dimensions is divided into 5 levels of perceived problems (level 1 = no problem, level 2 = slight problems, level 3 = moderate problems, level 4 = severe problems, level 5 = extreme problems). The participant selects an answer for each of the 5 dimensions considering the response that best matches his or her health "today." LOCF is defined as the participants who had a missing value or who stopped treatment at a specific time point had their last non-missing value carried forward.
Time Frame: Baseline, LOCF at Weeks 4, 8, 12, 16, 20, 24, 28, 32
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on Scale
Arm/Group | Esketamine Nasal Spray + Oral Antidepressant (AD) | Quetiapine Extended Release (XR) + Oral AD
Number analyzed (Participants) | 320 | 308
Units on Scale
  Week 4: number analyzed (Participants) | 318 | 306
  Week 4 | 0.177 (0.2354) | 0.124 (0.2280)
  Week 8 | 0.221 (0.2681) | 0.175 (0.2510)
  Week 12 | 0.247 (0.2552) | 0.187 (0.2523)
  Week 16 | 0.255 (0.2580) | 0.188 (0.2595)
  Week 20 | 0.261 (0.2600) | 0.187 (0.2590)
  Week 24 | 0.264 (0.2627) | 0.196 (0.2671)
  Week 28 | 0.266 (0.2739) | 0.195 (0.2664)
  Week 32 | 0.280 (0.2806) | 0.207 (0.2739)

19. Secondary Outcome: Change From Baseline in Participant-reported Health Status as Assessed by EQ-5D-5L Score: VAS
Description: Change from baseline in participant-reported health status as assessed by EQ-5D-5L Score: VAS was reported. The EQ-5D-5L is a standardized 2-part instrument for use as a measure of health outcome, primarily designed for self-completion by respondents. It essentially consists of the EQ-5D-5L descriptive system and the EQ-VAS. EQ-VAS self-rating records the respondent's own assessment of his/her overall health status at time of completion, on a scale of 0 (worst health you can imagine) to 100 (best health you can imagine). Positive change in score indicates improvement.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on Scale
Arm/Group | Esketamine Nasal Spray + Oral Antidepressant (AD) | Quetiapine Extended Release (XR) + Oral AD
Number analyzed (Participants) | 318 | 310
Units on Scale
  Week 4: number analyzed (Participants) | 317 | 308
  Week 4 | 13.3 (18.43) | 9.7 (17.83)
  Week 8: number analyzed (Participants) | 293 | 256
  Week 8 | 18.9 (19.84) | 16.1 (19.64)
  Week 12: number analyzed (Participants) | 280 | 238
  Week 12 | 20.9 (20.98) | 17.2 (20.73)
  Week 16: number analyzed (Participants) | 275 | 225
  Week 16 | 21.9 (20.14) | 20.2 (22.14)
  Week 20: number analyzed (Participants) | 267 | 215
  Week 20 | 22.3 (21.20) | 19.6 (21.59)
  Week 24: number analyzed (Participants) | 257 | 208
  Week 24 | 23.6 (20.95) | 21.8 (21.60)
  Week 28: number analyzed (Participants) | 251 | 205
  Week 28 | 25.2 (20.95) | 23.2 (22.11)
  Week 32: number analyzed (Participants) | 252 | 201
  Week 32 | 24.9 (21.65) | 24.5 (22.64)

20. Secondary Outcome: Change From Baseline in Participant-reported Health Status as Assessed by EQ-5D-5L Score: VAS at LOCF
Description: Change from baseline in participant-reported health status as assessed by EQ-5D-5L score: VAS at LOCF was reported. The EQ-5D-5L is a standardized 2-part instrument for use as a measure of health outcome, primarily designed for self-completion by respondents. It essentially consists of the EQ-5D-5L descriptive system and the EQ-VAS. EQ-VAS self-rating records the respondent's own assessment of his/her overall health status at time of completion, on a scale of 0 (worst health you can imagine) to 100 (best health you can imagine). Positive change in score indicates improvement. LOCF is defined as the participants who had a missing value or who stopped treatment at a specific time point had their last non-missing value carried forward.
Time Frame: Baseline, LOCF at Weeks 4, 8, 12, 16, 20, 24, 28, 32
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on Scale
Arm/Group | Esketamine Nasal Spray + Oral Antidepressant (AD) | Quetiapine Extended Release (XR) + Oral AD
Number analyzed (Participants) | 318 | 310
Units on Scale
  Week 4: number analyzed (Participants) | 317 | 308
  Week 4 | 13.3 (18.43) | 9.7 (17.83)
  Week 8 | 18.2 (19.94) | 14.0 (20.42)
  Week 12 | 19.4 (21.04) | 14.4 (21.19)
  Week 16 | 20.2 (20.37) | 16.1 (22.42)
  Week 20 | 20.4 (21.34) | 15.4 (22.19)
  Week 24 | 21.3 (21.34) | 16.9 (22.64)
  Week 28 | 21.9 (21.78) | 17.3 (23.10)
  Week 32 | 22.3 (22.47) | 18.0 (23.59)

21. Secondary Outcome: Change From Baseline in Participant-reported Work Productivity as Assessed by Work Productivity and Activity Impairment (WPAI): Depression Questionnaire
Description: Change from baseline in participant-reported work productivity as assessed by WPAI: depression questionnaire was reported. The WPAI-D questionnaire is a validated short instrument that assesses impairment in work and other regular activities over the past 7 days. The WPAI yields four types of scores: (a) Absenteeism (work time missed); (b) Presenteeism (impairment at work / reduced on-the-job effectiveness); (c) Work productivity loss (overall work impairment / absenteeism plus presenteeism); (d) Activity Impairment. The first three scores were derived only for respondents who were working (should be missing for non-working), but the last score was applicable for all respondents. Each score ranges from 0 to 100 with higher scores indicating greater impairment and less productivity.
Time Frame: Baseline, Weeks 4, 8, 12, 16, 20, 24, 28, 32
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Esketamine Nasal Spray + Oral Antidepressant (AD) | Quetiapine Extended Release (XR) + Oral AD
Number analyzed (Participants) | 310 | 307
Units on scale
  Absenteeism Week 4: number analyzed (Participants) | 115 | 112
  Absenteeism Week 4 | -11.95 (20.745) | -8.37 (25.790)
  Absenteeism Week 8: number analyzed (Participants) | 108 | 91
  Absenteeism Week 8 | -19.02 (30.205) | -13.62 (31.059)
  Absenteeism Week 12: number analyzed (Participants) | 106 | 72
  Absenteeism Week 12 | -21.87 (34.711) | -17.25 (31.340)
  Absenteeism Week 16: number analyzed (Participants) | 105 | 74
  Absenteeism Week 16 | -22.85 (33.023) | -14.24 (37.823)
  Absenteeism Week 20: number analyzed (Participants) | 102 | 78
  Absenteeism Week 20 | -27.88 (32.107) | -18.70 (35.310)
  Absenteeism Week 24: number analyzed (Participants) | 104 | 72
  Absenteeism Week 24 | -26.83 (32.909) | -21.03 (34.459)
  Absenteeism Week 28: number analyzed (Participants) | 97 | 73
  Absenteeism Week 28 | -27.16 (35.825) | -17.90 (31.254)
  Absenteeism Week 32: number analyzed (Participants) | 102 | 67
  Absenteeism Week 32 | -28.90 (32.066) | -16.68 (29.394)
  Presenteeism Week 4: number analyzed (Participants) | 120 | 115
  Presenteeism Week 4 | -21.75 (25.558) | -9.13 (21.948)
  Presenteeism Week 8: number analyzed (Participants) | 112 | 102
  Presenteeism Week 8 | -31.70 (25.144) | -16.86 (27.140)
  Presenteeism Week 12: number analyzed (Participants) | 108 | 87
  Presenteeism Week 12 | -35.46 (27.998) | -23.22 (29.942)
  Presenteeism Week 16: number analyzed (Participants) | 102 | 80
  Presenteeism Week 16 | -36.96 (28.556) | -24.50 (31.898)
  Presenteeism Week 20: number analyzed (Participants) | 99 | 82
  Presenteeism Week 20 | -39.80 (26.263) | -26.34 (33.389)
  Presenteeism Week 24: number analyzed (Participants) | 99 | 81
  Presenteeism Week 24 | -42.83 (27.332) | -31.60 (30.922)
  Presenteeism Week 28: number analyzed (Participants) | 100 | 79
  Presenteeism Week 28 | -43.00 (28.762) | -33.29 (34.445)
  Presenteeism Week 32: number analyzed (Participants) | 99 | 80
  Presenteeism Week 32 | -47.58 (26.691) | -33.88 (33.621)
  Work productivity loss Week 4: number analyzed (Participants) | 120 | 115
  Work productivity loss Week 4 | -20.94 (25.759) | -9.46 (23.374)
  Work productivity loss Week 8: number analyzed (Participants) | 112 | 102
  Work productivity loss Week 8 | -32.91 (26.244) | -18.21 (29.156)
  Work productivity loss Week 12: number analyzed (Participants) | 108 | 87
  Work productivity loss Week 12 | -36.68 (29.247) | -25.62 (35.135)
  Work productivity loss Week 16: number analyzed (Participants) | 102 | 80
  Work productivity loss Week 16 | -38.13 (30.490) | -24.50 (34.089)
  Work productivity loss Week 20: number analyzed (Participants) | 99 | 82
  Work productivity loss Week 20 | -41.11 (28.643) | -26.57 (32.885)
  Work productivity loss Week 24: number analyzed (Participants) | 99 | 81
  Work productivity loss Week 24 | -45.31 (29.000) | -30.63 (34.087)
  Work productivity loss Week 28: number analyzed (Participants) | 100 | 79
  Work productivity loss Week 28 | -44.40 (32.098) | -32.61 (33.836)
  Work productivity loss Week 32: number analyzed (Participants) | 99 | 80
  Work productivity loss Week 32 | -50.20 (29.176) | -35.48 (35.915)
  Activity Impairment Week 4: number analyzed (Participants) | 308 | 303
  Activity Impairment Week 4 | -20.29 (23.702) | -13.43 (20.846)
  Activity Impairment Week 8: number analyzed (Participants) | 287 | 254
  Activity Impairment Week 8 | -30.31 (27.410) | -24.25 (24.187)
  Activity Impairment Week 12: number analyzed (Participants) | 275 | 233
  Activity Impairment Week 12 | -33.96 (27.218) | -28.28 (25.555)
  Activity Impairment Week 16: number analyzed (Participants) | 270 | 221
  Activity Impairment Week 16 | -35.07 (27.291) | -30.95 (27.444)
  Activity Impairment Week 20: number analyzed (Participants) | 260 | 214
  Activity Impairment Week 20 | -33.88 (28.770) | -30.93 (27.698)
  Activity Impairment Week 24: number analyzed (Participants) | 248 | 206
  Activity Impairment Week 24 | -36.69 (29.742) | -36.84 (27.000)
  Activity Impairment Week 28: number analyzed (Participants) | 244 | 202
  Activity Impairment Week 28 | -40.00 (29.828) | -37.62 (28.500)
  Activity Impairment Week 32: number analyzed (Participants) | 245 | 196
  Activity Impairment Week 32 | -41.92 (30.299) | -39.59 (27.190)

22. Secondary Outcome: Change From Baseline in Participant-reported Work Productivity as Assessed by WPAI: Depression Questionnaire at LOCF
Description: Change from baseline in participant-reported work productivity as assessed by WPAI: depression questionnaire at LOCF was reported. The WPAI-D questionnaire is a validated short instrument that assesses impairment in work and other regular activities over the past 7 days. The WPAI yields four types of scores: (a) Absenteeism (work time missed); (b) Presenteeism (impairment at work / reduced on-the-job effectiveness); (c) Work productivity loss (overall work impairment / absenteeism plus presenteeism); (d) Activity Impairment. The first three scores were derived only for respondents who were working (should be missing for non-working), but the last score was applicable for all respondents. Each score ranges from 0 to 100 with higher scores indicating greater impairment and less productivity. LOCF is defined as the participants who had a missing value or who stopped treatment at a specific time point had their last non-missing value carried forward.
Time Frame: Baseline, LOCF at Weeks 4, 8, 12, 16, 20, 24, 28, 32
Population: The FAS included all randomized participants. Here, 'N' (number of participants analyzed) signifies participants evaluable for this outcome measure. Here, 'n' (number analyzed) signifies participants evaluable for this outcome measure at specified time points. LOCF was applied only for participants whose questionnaire was completely missing. No LOCF imputation was done on partially completed questionnaire.
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Esketamine Nasal Spray + Oral Antidepressant (AD) | Quetiapine Extended Release (XR) + Oral AD
Number analyzed (Participants) | 310 | 307
Units on scale
  Absenteeism Week 4: number analyzed (Participants) | 115 | 112
  Absenteeism Week 4 | -11.95 (20.745) | -8.37 (25.790)
  Absenteeism Week 8: number analyzed (Participants) | 120 | 107
  Absenteeism Week 8 | -18.28 (29.417) | -12.38 (30.369)
  Absenteeism Week 12: number analyzed (Participants) | 120 | 103
  Absenteeism Week 12 | -20.23 (33.590) | -15.17 (31.835)
  Absenteeism Week 16: number analyzed (Participants) | 122 | 107
  Absenteeism Week 16 | -21.35 (31.806) | -14.14 (37.534)
  Absenteeism Week 20: number analyzed (Participants) | 124 | 114
  Absenteeism Week 20 | -25.45 (31.628) | -16.04 (37.769)
  Absenteeism Week 24: number analyzed (Participants) | 126 | 111
  Absenteeism Week 24 | -24.41 (32.403) | -16.28 (37.672)
  Absenteeism Week 28: number analyzed (Participants) | 122 | 114
  Absenteeism Week 28 | -23.88 (34.623) | -14.14 (35.849)
  Absenteeism Week 32: number analyzed (Participants) | 128 | 108
  Absenteeism Week 32 | -26.10 (31.903) | -13.90 (36.104)
  Presenteeism Week 4: number analyzed (Participants) | 120 | 115
  Presenteeism Week 4 | -21.75 (25.558) | -9.13 (21.948)
  Presenteeism Week 8: number analyzed (Participants) | 127 | 122
  Presenteeism Week 8 | -29.45 (26.437) | -14.84 (27.067)
  Presenteeism Week 12: number analyzed (Participants) | 129 | 125
  Presenteeism Week 12 | -33.57 (28.745) | -17.44 (29.997)
  Presenteeism Week 16: number analyzed (Participants) | 130 | 128
  Presenteeism Week 16 | -35.00 (29.075) | -19.84 (31.322)
  Presenteeism Week 20: number analyzed (Participants) | 130 | 128
  Presenteeism Week 20 | -36.08 (28.598) | -21.41 (32.862)
  Presenteeism Week 24: number analyzed (Participants) | 131 | 128
  Presenteeism Week 24 | -36.87 (29.641) | -22.19 (32.189)
  Presenteeism Week 28: number analyzed (Participants) | 131 | 128
  Presenteeism Week 28 | -37.40 (30.924) | -23.83 (34.757)
  Presenteeism Week 32: number analyzed (Participants) | 131 | 128
  Presenteeism Week 32 | -40.53 (30.700) | -23.44 (35.526)
  Work productivity loss Week 4: number analyzed (Participants) | 120 | 115
  Work productivity loss Week 4 | -20.94 (25.759) | -9.46 (23.374)
  Work productivity loss Week 8: number analyzed (Participants) | 127 | 122
  Work productivity loss Week 8 | -30.59 (26.789) | -15.35 (30.059)
  Work productivity loss Week 12: number analyzed (Participants) | 129 | 125
  Work productivity loss Week 12 | -34.46 (29.333) | -19.27 (33.905)
  Work productivity loss Week 16: number analyzed (Participants) | 130 | 128
  Work productivity loss Week 16 | -36.35 (30.531) | -20.75 (33.545)
  Work productivity loss Week 20: number analyzed (Participants) | 130 | 128
  Work productivity loss Week 20 | -37.59 (30.354) | -22.58 (34.117)
  Work productivity loss Week 24: number analyzed (Participants) | 131 | 128
  Work productivity loss Week 24 | -39.02 (31.482) | -22.54 (34.635)
  Work productivity loss Week 28: number analyzed (Participants) | 131 | 128
  Work productivity loss Week 28 | -39.09 (33.271) | -23.85 (35.152)
  Work productivity loss Week 32: number analyzed (Participants) | 132 | 128
  Work productivity loss Week 32 | -43.42 (32.638) | -24.89 (37.870)
  Activity Impairment Week 4: number analyzed (Participants) | 308 | 303
  Activity Impairment Week 4 | -20.29 (23.702) | -13.43 (20.846)
  Activity Impairment Week 8: number analyzed (Participants) | 310 | 306
  Activity Impairment Week 8 | -28.84 (27.412) | -20.39 (24.599)
  Activity Impairment Week 12: number analyzed (Participants) | 310 | 306
  Activity Impairment Week 12 | -31.10 (27.778) | -22.81 (26.264)
  Activity Impairment Week 16 | -31.84 (28.413) | -23.68 (28.014)
  Activity Impairment Week 20 | -30.84 (29.983) | -23.62 (28.185)
  Activity Impairment Week 24 | -32.45 (31.207) | -26.71 (28.821)
  Activity Impairment Week 28 | -34.87 (31.804) | -27.07 (29.965)
  Activity Impairment Week 32 | -36.65 (32.357) | -28.40 (29.930)

23. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: An AE is any untoward medical occurrence in a participant participating in a clinical study that does not necessarily have a causal relationship with the pharmaceutical/ biological agent under study. TEAEs were those events if they started after administration of the first dose until 14 days after the last dose of study medication for other TEAEs except serious; and first dose until 30 days after the last dose of study medication for serious TEAEs.
Time Frame: Up to Week 35
Population: The safety analysis set included all randomized participants who received at least 1 dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Esketamine Nasal Spray + Oral Antidepressant (AD) | Quetiapine Extended Release (XR) + Oral AD
Number analyzed (Participants) | 334 | 336
Participants | 307 | 262

24. Secondary Outcome: Number of Participants With TEAEs of Special Interest
Description: Number of participants with TEAEs of special interest were reported. It included significant TEAEs that were judged to be of special interest because of clinical importance, known or suspected class effects, or based on nonclinical signals. Events such as sedation, depersonalization/derealization disorder, depression suicidal, aggression, allergic cystitis, cholestasis and jaundice of hepatic origin, and many more were considered as TEAEs of special interest.
Time Frame: Up to Week 35
Population: The safety analysis set included all randomized participants who received at least 1 dose of any study intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Esketamine Nasal Spray + Oral Antidepressant (AD) | Quetiapine Extended Release (XR) + Oral AD
Number analyzed (Participants) | 334 | 336
Participants | 223 | 140

25. Secondary Outcome: Number of Participants With Suicidal Ideation or Behavior as Assessed by Columbia-Suicide Severity Rating Scale (C-SSRS) Score
Description: Number of participants with suicidal ideation or behavior as assessed by C-SSRS score was reported. The C-SSRS is an assessment tool that evaluates suicidal ideation and behavior. Suicidal ideation consists of 5 items: wish to be dead, non-specific active suicidal thoughts, active suicidal ideation with any methods (not plan) without intention to act, active suicidal ideation with some intent to act without specific plan, and active suicidal ideation with specific plan and intent. Suicidal behavior consists of 5 items: preparatory acts or behavior, aborted attempt, interrupted attempt, actual attempt (non-fatal), and completed suicide. The maximum score (from the 10 categories) assigned for each participant was summarized into one of three broad categories: No suicidal ideation or behavior (0), Suicidal ideation (1 - 5), Suicidal behavior (6 - 10). Total score ranges from 1 to 10. Higher scores indicate more severe suicidal ideation and behavior.
Time Frame: Weeks 1, 2, 3, 4, 8, 12, 16, 20, 24, 28, 32
Population: The safety analysis set included all randomized participants who received at least 1 dose of any study intervention. Here, 'N' (number of participants analyzed) signifies participants evaluable for this outcome measure. Here, 'n' (number analyzed) signifies participants evaluable for this outcome measure at specified time points.
Measure: Count of Participants; unit: Participants
Arm/Group | Esketamine Nasal Spray + Oral Antidepressant (AD) | Quetiapine Extended Release (XR) + Oral AD
Number analyzed (Participants) | 317 | 295
Participants
  Suicidal Ideation Week 1: number analyzed (Participants) | 277 | 282
  Suicidal Ideation Week 1 | 22 | 25
  Suicidal Behavior Week 1: number analyzed (Participants) | 277 | 282
  Suicidal Behavior Week 1 | 0 | 0
  Suicidal Ideation Week 2: number analyzed (Participants) | 278 | 274
  Suicidal Ideation Week 2 | 21 | 32
  Suicidal Behavior Week 2: number analyzed (Participants) | 278 | 274
  Suicidal Behavior Week 2 | 0 | 1
  Suicidal Ideation Week 3: number analyzed (Participants) | 271 | 265
  Suicidal Ideation Week 3 | 19 | 17
  Suicidal Behavior Week 3: number analyzed (Participants) | 271 | 265
  Suicidal Behavior Week 3 | 0 | 0
  Suicidal Ideation Week 4 | 22 | 27
  Suicidal Behavior Week 4 | 0 | 0
  Suicidal Ideation Week 8: number analyzed (Participants) | 300 | 265
  Suicidal Ideation Week 8 | 21 | 18
  Suicidal Behavior Week 8: number analyzed (Participants) | 300 | 265
  Suicidal Behavior Week 8 | 0 | 0
  Suicidal Ideation Week 12: number analyzed (Participants) | 286 | 239
  Suicidal Ideation Week 12 | 13 | 14
  Suicidal Behavior Week 12: number analyzed (Participants) | 286 | 239
  Suicidal Behavior Week 12 | 0 | 0
  Suicidal Ideation Week 16: number analyzed (Participants) | 280 | 229
  Suicidal Ideation Week 16 | 12 | 12
  Suicidal Behavior Week 16: number analyzed (Participants) | 280 | 229
  Suicidal Behavior Week 16 | 1 | 1
  Suicidal Ideation Week 20: number analyzed (Participants) | 270 | 218
  Suicidal Ideation Week 20 | 15 | 14
  Suicidal Behavior Week 20: number analyzed (Participants) | 270 | 218
  Suicidal Behavior Week 20 | 0 | 0
  Suicidal Ideation Week 24: number analyzed (Participants) | 260 | 213
  Suicidal Ideation Week 24 | 14 | 9
  Suicidal Behavior Week 24: number analyzed (Participants) | 260 | 213
  Suicidal Behavior Week 24 | 0 | 0
  Suicidal Ideation Week 28: number analyzed (Participants) | 255 | 208
  Suicidal Ideation Week 28 | 8 | 5
  Suicidal Behavior Week 28: number analyzed (Participants) | 255 | 208
  Suicidal Behavior Week 28 | 0 | 0
  Suicidal Ideation Week 32: number analyzed (Participants) | 250 | 203
  Suicidal Ideation Week 32 | 7 | 4
  Suicidal Behavior Week 32: number analyzed (Participants) | 250 | 203
  Suicidal Behavior Week 32 | 0 | 1

ADVERSE EVENTS:
Time Frame: All-cause mortality and serious adverse events: until 30 days after last dose (up to Week 35); other AEs: until 14 days after last dose (up to Week 33)
Description: The safety analysis set included all randomized participants who received at least 1 dose of any study intervention.
Arm/Group | Esketamine Nasal Spray + Oral Antidepressant (AD) | Quetiapine Extended Release (XR) + Oral AD
All-Cause Mortality (participants affected / at risk) | 1/334 | 1/336
Serious Adverse Events (participants affected / at risk) | 19/334 | 17/336
Other Adverse Events (participants affected / at risk) | 289/334 | 216/336
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Esketamine Nasal Spray + Oral Antidepressant (AD) (N=334) | Quetiapine Extended Release (XR) + Oral AD (N=336)
Lymphadenopathy mediastinal (Blood and lymphatic system disorders) | 0 | 1
Acute coronary syndrome (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Retinal detachment (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Death (General disorders) | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1
COVID-19 (Infections and infestations) | 1 | 0
Cystitis (Infections and infestations) | 0 | 1
Pilonidal disease (Infections and infestations) | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Generalised tonic-clonic seizure (Nervous system disorders) | 0 | 1
Alcoholism (Psychiatric disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 2
Conversion disorder (Psychiatric disorders) | 0 | 1
Depression (Psychiatric disorders) | 2 | 3
Major depression (Psychiatric disorders) | 1 | 1
Somatic symptom disorder (Psychiatric disorders) | 2 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 3
Suicide attempt (Psychiatric disorders) | 2 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Esketamine Nasal Spray + Oral Antidepressant (AD) (N=334) | Quetiapine Extended Release (XR) + Oral AD (N=336)
Vertigo (Ear and labyrinth disorders) | 63 | 3
Vision blurred (Eye disorders) | 21 | 3
Dry mouth (Gastrointestinal disorders) | 3 | 22
Nausea (Gastrointestinal disorders) | 98 | 12
Vomiting (Gastrointestinal disorders) | 36 | 5
Fatigue (General disorders) | 19 | 34
COVID-19 (Infections and infestations) | 24 | 29
Nasopharyngitis (Infections and infestations) | 21 | 11
Blood pressure increased (Investigations) | 28 | 4
Weight increased (Investigations) | 9 | 42
Back pain (Musculoskeletal and connective tissue disorders) | 17 | 9
Dizziness (Nervous system disorders) | 156 | 28
Dysgeusia (Nervous system disorders) | 40 | 1
Headache (Nervous system disorders) | 82 | 43
Hypoaesthesia (Nervous system disorders) | 19 | 1
Paraesthesia (Nervous system disorders) | 37 | 2
Sedation (Nervous system disorders) | 22 | 29
Somnolence (Nervous system disorders) | 50 | 78
Confusional state (Psychiatric disorders) | 20 | 1
Dissociation (Psychiatric disorders) | 94 | 2

LIMITATIONS AND CAVEATS:
To minimize potential bias, the Montgomery-Asberg Depression Rating Scale (MADRS) was performed by an independent on-site rater who was blinded to the participant's treatment, and who was not involved in any other study assessments or treatment decisions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.

DOCUMENTS (2):
  • Study Protocol (2020-10-08): https://cdn.clinicaltrials.gov/large-docs/21/NCT04338321/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-12): https://cdn.clinicaltrials.gov/large-docs/21/NCT04338321/SAP_001.pdf